CLINICAL TRIAL: NCT04823650
Title: Low-Interventional Study to Record Gait and Physical Activity Using ActiGraph Devices in Children Ages 3-17.
Brief Title: Monitoring Activity And Gait In Children
Acronym: MAGIC
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: X9001263; MAGIC (Other: Alias Study Number)
Record Dates: First submitted 2021-03-18; First posted 2021-04-01 (Actual); Results first posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Child, Preschool; Child; Adolescent
Keywords: COHORT A :; Gait; Activity; Actigraphy; COHORT B:; Sleep
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (3):
- Ages 3-5: COHORT A and B
  Interventions: Device: COHORT A: Actigraph; Device: Panoramic Bracelet and GENEActiv
- Ages 6-11: COHORT A and B
  Interventions: Device: COHORT A: Actigraph; Device: Panoramic Bracelet and GENEActiv
- Ages 12-17: COHORT A and B
  Interventions: Device: COHORT A: Actigraph; Device: Panoramic Bracelet and GENEActiv

INTERVENTIONS:
Device: COHORT A: Actigraph — The ActiGraph CentrePoint Insight Watch is a small worn activity monitor designed for documenting physical movement associated with applications in physiological monitoring.
Device: Panoramic Bracelet and GENEActiv — Panoramic Bracelet:
  The Panoramic Digital Health Bracelet is a wearable inertial measurement unit "intended for use by researchers and healthcare professionals for high frequency or continuous collection of physical data in home and professional healthcare settings during research studies." It includes a 3 axis accelerometer and gyroscope, as well as magnetometer, pressure, and temperature sensors. The bracelet has no interface or screen for participants to interact with.
  GENEActiv:
  The GENEActiv device is a wearable inertial measurement unit "designed for public health research and clinical trials." The device is a circular unit with attachable wrist-bands, and has no interface or screen for participants to interact with. The GENEActiv device is FDA 510(k) exempt. The device records acceleration data and can collect data remotely for up to 1 month.

SUMMARY:
COHORT A: To study whether a digital health tool called Actigraph can be used to collect information on gait and physical activity in healthy children aged 3-17. The study will be conducted at the Pfizer Innovation Research Laboratory (PfIRe Lab) in Cambridge MA. In the lab at the first visit, we will ask participants to do activities such as walking on different surfaces as well as to roll a dice and move between different activity stations. Children will wear 2 Actigraph devices, one as a watch and one as a belt. They will then go home and do usual daily activities while answering a brief daily activity diary for approximately 2 weeks. The conclusion of the study will be over the telephone and include questions on the comfort and wearability of the device. The analysis of gait and physical activity as well as adherence and wearability will be looked across three different age groups 3-5, 6-11, and 12-17.

COHORT B: Cohort B of the study aims to evaluate the feasibility of the Panoramic Bracelet and associated algorithms such as SleepPy and GaitPy compared to the GENEActiv device and to evaluate the comfort and wearability of the Panoramic Bracelet. The results of this study will enable the use of novel devices in future clinical trials measuring scratch and sleep. . In the lab at the first visit, we will ask participants to do activities such as walking on different surfaces as well as to roll a dice and move between different activity stations. They will then go home and do usual daily activities while wearing both devices in the same wrist at different times stipulated in the protocol, answering a brief daily activity and sleep diary for approximately 2 weeks. Cohort B includes questions on the comfort and wearability of the Panoramic device on Day 7 approximately. The conclusion of the study will be over the telephone.The analysis will be looked across three different age groups 3-5, 6-11, and 12-17

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory
* No significant health problems that would impair the completion of the physical activity tasks, does not carry any diagnosis of developmental delay and/or significant co-morbid medical conditions as determined by a medically qualified individual during medical history review

Exclusion Criteria:

* Participation in other studies involving digital devices within 1 week and/or treatment with an investigational drug (Phases 1-4) within 30 days or 5 half-lives before the current study begins and/or during study participation.
* Participants with implanted medical devices.
* Minor participants who reach the age of majority during the study, as recognized under local law.
* Any medical or psychiatric condition that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* Participants with known allergies to components as specified by device manufacturer if applicable (eg, plastic, stainless steel and silicone).

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy children and adolescents aged 3-17.
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2024-10-28 (Actual); Study Completion 2024-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Innovation Research, PfIRe, Lab, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Di J, Tuttle PG, Adamowicz L, Lin W, Zhang H, Psaltos D, Selig J, Bai J, Karahanoglu FI, Sheriff P, Seelam V, Williams B, Ghafoor S, Demanuele C, Santamaria M, Cai X. Monitoring Activity and Gait in Children (MAGIC) using digital health technologies. Pediatr Res. 2024 Aug;96(3):750-758. doi: 10.1038/s41390-024-03147-x. Epub 2024 Mar 21. PMID 38514860
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=X9001263

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In this observational study, healthy pediatric participants (aged 3-17) were enrolled in 2 cohorts: Cohort A and B. A total of 87 participants (Cohort A: 40 and Cohort B: 47) were screened and enrolled in the study. No intervention was administered during this study.
Groups:
- Cohort A: Participants Aged 3-5 Years: Participants aged 3 to 5 years wore the ActiGraph CenterPoint Insight Watch on the non-dominant wrist (worn continuously) and lumbar region (worn after waking up in the morning and removed while sleeping at night or nap during daytime) for approximately 15 days (+ 3 days). Participants wore the Ambulatory Parkinson's Disease Monitoring System (APDM) Opal sensors on each wrist, chest, lumbar, and above each shoe, only on Day 1.
- Cohort A: Participants Aged 6-11 Years: Participants aged 6 to 11 years wore the ActiGraph CenterPoint Insight Watch on the non-dominant wrist (worn continuously) and lumbar region (worn after waking up in the morning and removed while sleeping at night or nap during daytime) for approximately 15 days (+ 3 days). Participants wore the APDM Opal sensors on each wrist, chest, lumbar, and above each shoe, only on Day 1.
- Cohort A: Participants Aged 12-17 Years: Participants aged 12 to 17 years wore the ActiGraph CenterPoint Insight Watch on the non-dominant wrist (worn continuously) and lumbar region (worn after waking up in the morning and removed while sleeping at night or nap during daytime) for approximately 15 days (+ 3 days). Participants wore the APDM Opal sensors on each wrist, chest, lumbar, and above each shoe, only on Day 1.
- Cohort B: Participants Aged 3-5 Years: Participants aged 3 to 5 years wore the Panoramic Digital Health Bracelet on the non-dominant wrist for approximately 15 days (+ 3 days). GENEActiv device was also worn on the same non-dominant wrist from Day 7 (+ 2 days) to Day 15 (+ 2 days). Participants wore the APDM Opal sensors on each wrist, chest, lumbar, and above each shoe, only on Day 1.
- Cohort B: Participants Aged 6-11 Years: Participants aged 6 to 11 years wore the Panoramic Digital Health Bracelet on the non-dominant wrist for approximately 15 days (+ 3 days). GENEActiv device was also worn on the same non-dominant wrist from Day 7 (+ 2 days) to Day 15 (+ 2 days). Participants wore the APDM Opal sensors on each wrist, chest, lumbar, and above each shoe, only on Day 1.
- Cohort B: Participants Aged 12-17 Years: Participants aged 12 to 17 years wore the Panoramic Digital Health Bracelet on the non-dominant wrist for approximately 15 days (+ 3 days). GENEActiv device was also worn on the same non-dominant wrist from Day 7 (+ 2 days) to Day 15 (+ 2 days). Participants wore the APDM Opal sensors on each wrist, chest, lumbar, and above each shoe, only on Day 1.
Period: Overall Study
Arm/Group | Cohort A: Participants Aged 3-5 Years | Cohort A: Participants Aged 6-11 Years | Cohort A: Participants Aged 12-17 Years | Cohort B: Participants Aged 3-5 Years | Cohort B: Participants Aged 6-11 Years | Cohort B: Participants Aged 12-17 Years
Started | 13 | 14 | 13 | 13 | 17 | 17
Completed | 13 | 14 | 13 | 13 | 16 | 17
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: Participants Aged 3-5 Years | Cohort A: Participants Aged 6-11 Years | Cohort A: Participants Aged 12-17 Years | Cohort B: Participants Aged 3-5 Years | Cohort B: Participants Aged 6-11 Years | Cohort B: Participants Aged 12-17 Years | Total
Number analyzed (Participants) | 13 | 14 | 13 | 13 | 17 | 17 | 87
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Here, 'Number Analyzed' signifies number of participants evaluable for the specified rows.
  Years
    Cohort A: number analyzed (Participants) | 13 | 14 | 13 | 0 | 0 | 0 | 40
    Cohort A | 4.38 (0.65) | 9.00 (1.80) | 14.77 (1.59) |  |  |  | 9.38 (4.48)
    Cohort B: number analyzed (Participants) | 0 | 0 | 0 | 13 | 17 | 17 | 47
    Cohort B |  |  |  | 4.00 (0.82) | 8.53 (1.62) | 13.94 (1.68) | 9.23 (4.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 9 | 8 | 8 | 11 | 49
  Male | 6 | 8 | 4 | 5 | 9 | 6 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 2 | 0 | 4 | 0 | 9
  Not Hispanic or Latino | 11 | 11 | 11 | 13 | 13 | 17 | 76
  Unknown or Not Reported | 0 | 2 | 0 | 0 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 3 | 5 | 1 | 3 | 0 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1 | 1 | 0 | 3
  White | 8 | 10 | 8 | 8 | 12 | 16 | 62
  More than one race | 1 | 1 | 0 | 3 | 1 | 1 | 7
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Cohort A: Gait Speed Measured by APDM, GAITRite Walkway and ActiGraph Devices for Walk at Natural, Slow and Fast Speed Tasks
Description: Gait speed was the time taken to walk a specified distance. Participants had to walk on GAITRite walkway (20 feet*3) wearing ActiGraph and APDM devices at participant's natural speed and at varied speeds. Natural speed was participant's self-chosen pace for 3 rounds. Varied speeds included participant's self-chosen slow pace ("Walk slow") and fast pace ("Walk fast") for 3 rounds. Raw accelerometry data collected by ActiGraph devices (comparator) was processed by the GaitPy algorithm to generate gait quality metrics (lumbar position). Gait metrics data was directly extracted from GAITRite walkway and APDM sensors (reference).
Time Frame: Up to 20 minutes on Day 1
Population: FAS included all participants who had a signed and dated informed consent document, had assented to the study and were enrolled in the study. Here, 'Number Analyzed' signifies number of participants evaluable for the specified rows. The outcome measure was planned to be evaluated only for Cohort A.
Measure: Mean (Standard Deviation); unit: Meters per second
Arm/Group | Cohort A: Participants Aged 3-5 Years | Cohort A: Participants Aged 6-11 Years | Cohort A: Participants Aged 12-17 Years
Number analyzed (Participants) | 13 | 14 | 13
Meters per second
  ActiGraph: Natural Speed | 0.83 (0.192) | 1.00 (0.142) | 1.04 (0.174)
  GAITRite: Natural Speed | 0.93 (0.234) | 1.13 (0.127) | 1.21 (0.177)
  APDM: Natural Speed | 0.81 (0.213) | 1.02 (0.119) | 1.10 (0.171)
  ActiGraph: Fast Speed | 1.03 (0.231) | 1.22 (0.129) | 1.30 (0.115)
  GAITRite: Fast Speed | 1.32 (0.268) | 1.49 (0.252) | 1.56 (0.161)
  APDM: Fast Speed: number analyzed (Participants) | 11 | 14 | 13
  APDM: Fast Speed | 1.00 (0.218) | 1.36 (0.247) | 1.43 (0.139)
  ActiGraph: Slow Speed: number analyzed (Participants) | 13 | 12 | 13
  ActiGraph: Slow Speed | 0.56 (0.150) | 0.58 (0.173) | 0.64 (0.173)
  GAITRite: Slow Speed | 0.57 (0.164) | 0.54 (0.151) | 0.75 (0.204)
  APDM: Slow Speed | 0.49 (0.159) | 0.45 (0.153) | 0.66 (0.196)
Statistical Analysis 1: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Natural Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.79, 95% CI 2-sided [-0.16 to 0.95] — Agreement between two devices' measurements was assessed by the intraclass correlation coefficient as: <= 0.4 (poor), 0.4 to 0.59 (moderate), 0.6 to 0.74 (good), and 0.75 to 1 (excellent) agreement
Statistical Analysis 2: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Natural Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.606, 95% CI 2-sided [-0.10 to 0.91] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Natural Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.637, 95% CI 2-sided [-0.05 to 0.92] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Natural Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.741, 95% CI 2-sided [0.33 to 0.91] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Natural Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.88, 95% CI 2-sided [0.65 to 0.96] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Natural Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.892, 95% CI 2-sided [-0.16 to 0.98] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Natural Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.77, 95% CI 2-sided [0.36 to 0.93] — Agreement between devices' measurements was assessed by the intraclass correlation coefficient as: <= 0.4 (poor), 0.4 to 0.59 (moderate), 0.6 to 0.74 (good), and 0.75 to 1 (excellent) agreement
Statistical Analysis 8: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Natural Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.715, 95% CI 2-sided [-0.08 to 0.94] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 9: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Natural Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.767, 95% CI 2-sided [-0.04 to 0.96] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 10: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Fast Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.428, 95% CI 2-sided [-0.17 to 0.84] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Fast Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.335, 95% CI 2-sided [-0.16 to 0.77] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Fast Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.273, 95% CI 2-sided [-0.07 to 0.74] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Fast Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.854, 95% CI 2-sided [0.58 to 0.95] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 14: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Fast Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.537, 95% CI 2-sided [-0.13 to 0.85] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 15: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Fast Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.536, 95% CI 2-sided [-0.15 to 0.89] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 16: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Fast Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.527, 95% CI 2-sided [-0.10 to 0.87] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 17: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Fast Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.574, 95% CI 2-sided [-0.10 to 0.88] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 18: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Fast Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.454, 95% CI 2-sided [-0.05 to 0.85] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 19: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Slow Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.834, 95% CI 2-sided [0.54 to 0.95] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 20: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Slow Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.317, 95% CI 2-sided [-0.27 to 0.72] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 21: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Slow Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.789, 95% CI 2-sided [-0.18 to 0.96] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 22: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Slow Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.737, 95% CI 2-sided [0.09 to 0.92] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 23: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Slow Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.3, 95% CI 2-sided [-0.19 to 0.69] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 24: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Slow Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.936, 95% CI 2-sided [0.81 to 0.98] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 25: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Slow Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.82, 95% CI 2-sided [0.42 to 0.95] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 26: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Slow Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.521, 95% CI 2-sided [0.19 to 0.79] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 27: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Slow Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.871, 95% CI 2-sided [-0.09 to 0.98] — [estimate comment as in outcome 1, analysis 7]

2. Primary Outcome: Cohort A: Double Support Duration Measured by APDM, GAITRite Walkway and ActiGraph Devices for Walk at Natural, Slow and Fast Speed Tasks
Description: Double support time referred to the phase during walking when both feet were in contact with the ground. Participants had to walk on GAITRite walkway (20 feet*3) wearing ActiGraph and APDM devices at participant's natural speed and at varied speeds. Natural speed was participant's self-chosen pace for 3 rounds. Varied speeds included participant's self-chosen slow pace ("Walk slow") and fast pace ("Walk fast") for 3 rounds. Raw accelerometry data collected by ActiGraph devices (comparator) was processed by the GaitPy algorithm to generate gait quality metrics (lumbar position). Gait metrics data was directly extracted from GAITRite walkway and APDM sensors (reference).
Time Frame: Up to 20 minutes on Day 1
Population: Full Analysis Set (FAS) included all participants who had a signed and dated informed consent document, had assented to the study and were enrolled in the study. Here, 'Number Analyzed' signifies number of participants evaluable for the specified rows. The outcome measure was planned to be evaluated only for Cohort A.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Cohort A: Participants Aged 3-5 Years | Cohort A: Participants Aged 6-11 Years | Cohort A: Participants Aged 12-17 Years
Number analyzed (Participants) | 13 | 14 | 13
Seconds
  ActiGraph: Natural Speed | 0.26 (0.031) | 0.27 (0.029) | 0.30 (0.022)
  GAITRite: Natural Speed | 0.28 (0.096) | 0.26 (0.053) | 0.31 (0.049)
  APDM: Natural Speed | 0.22 (0.081) | 0.17 (0.033) | 0.21 (0.048)
  ActiGraph: Fast Speed | 0.23 (0.020) | 0.24 (0.028) | 0.27 (0.020)
  GAITRite: Fast Speed | 0.18 (0.048) | 0.20 (0.057) | 0.24 (0.042)
  APDM: Fast Speed: number analyzed (Participants) | 11 | 12 | 13
  APDM: Fast Speed | 0.16 (0.027) | 0.13 (0.031) | 0.14 (0.039)
  ActiGraph: Slow Speed | 0.29 (0.024) | 0.32 (0.039) | 0.32 (0.034)
  GAITRite: Slow Speed | 0.45 (0.155) | 0.60 (0.192) | 0.53 (0.139)
  APDM: Slow Speed | 0.36 (0.150) | 0.41 (0.144) | 0.38 (0.126)
Statistical Analysis 1: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Natural Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.548, 95% CI 2-sided [0.02 to 0.84] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Natural Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.731, 95% CI 2-sided [0.35 to 0.91] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Natural Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.623, 95% CI 2-sided [0.14 to 0.87] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Natural Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.491, 95% CI 2-sided [-0.11 to 0.82] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Natural Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.136, 95% CI 2-sided [-0.01 to 0.52] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Natural Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.157, 95% CI 2-sided [-0.04 to 0.59] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Natural Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.649, 95% CI 2-sided [0.17 to 0.88] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 8: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Natural Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.259, 95% CI 2-sided [-0.04 to 0.71] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 9: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Natural Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.242, 95% CI 2-sided [-0.04 to 0.70] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 10: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Fast Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.24, 95% CI 2-sided [-0.18 to 0.66] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Fast Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.481, 95% CI 2-sided [-0.21 to 0.83] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Fast Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.31, 95% CI 2-sided [-0.19 to 0.72] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Fast Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.096, 95% CI 2-sided [-0.07 to 0.46] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 14: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Fast Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.1, 95% CI 2-sided [-0.01 to 0.44] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 15: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Fast Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.058, 95% CI 2-sided [-0.02 to 0.35] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 16: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Fast Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.206, 95% CI 2-sided [-0.08 to 0.59] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 17: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Fast Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.247, 95% CI 2-sided [-0.05 to 0.70] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 18: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Fast Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.127, 95% CI 2-sided [-0.03 to 0.53] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 19: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Slow Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = -0.031, 95% CI 2-sided [-0.25 to 0.34] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 20: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Slow Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.004, 95% CI 2-sided [-0.13 to 0.27] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 21: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Slow Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = -0.085, 95% CI 2-sided [-0.21 to 0.21] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 22: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Slow Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = -0.077, 95% CI 2-sided [-0.50 to 0.44] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 23: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Slow Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.063, 95% CI 2-sided [-0.31 to 0.50] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 24: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Slow Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = -0.248, 95% CI 2-sided [-0.62 to 0.29] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 25: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Slow Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.331, 95% CI 2-sided [-0.02 to 0.69] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 26: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Slow Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.217, 95% CI 2-sided [-0.08 to 0.59] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 27: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Slow Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.169, 95% CI 2-sided [-0.07 to 0.52] — [estimate comment as in outcome 1, analysis 7]

3. Primary Outcome: Cohort A: Single Limb Support Duration Measured by APDM, GAITRite Walkway and ActiGraph Devices for Walk at Natural, Slow and Fast Speed Tasks
Description: Single support time referred to the time when only one limb was in contact with the ground. Participants had to walk on GAITRite walkway (20 feet*3) wearing ActiGraph and APDM devices at participant's natural speed and at varied speeds. Natural speed was participant's self-chosen pace for 3 rounds. Varied speeds included participant's self-chosen slow pace ("Walk slow") and fast pace ("Walk fast") for 3 rounds. Raw accelerometery data collected by ActiGraph devices (comparator) was processed by the GaitPy algorithm to generate gait quality metrics (lumbar position). Gait metrics data was directly extracted from GAITRite walkway and APDM sensors (reference).
Time Frame: Up to 20 minutes on Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Cohort A: Participants Aged 3-5 Years | Cohort A: Participants Aged 6-11 Years | Cohort A: Participants Aged 12-17 Years
Number analyzed (Participants) | 13 | 14 | 13
Seconds
  ActiGraph: Natural Speed | 0.36 (0.054) | 0.38 (0.050) | 0.42 (0.028)
  GAITRite: Natural Speed | 0.36 (0.034) | 0.37 (0.037) | 0.40 (0.027)
  APDM: Natural Speed | 0.39 (0.045) | 0.42 (0.042) | 0.46 (0.022)
  ActiGraph: Fast Speed | 0.31 (0.036) | 0.34 (0.042) | 0.37 (0.026)
  GAITRite: Fast Speed | 0.30 (0.031) | 0.34 (0.039) | 0.38 (0.029)
  APDM: Fast Speed: number analyzed (Participants) | 11 | 14 | 13
  APDM: Fast Speed | 0.36 (0.027) | 0.39 (0.042) | 0.42 (0.024)
  ActiGraph: Slow Speed | 0.47 (0.080) | 0.59 (0.140) | 0.58 (0.123)
  GAITRite: Slow Speed | 0.43 (0.058) | 0.51 (0.074) | 0.48 (0.045)
  APDM: Slow Speed | 0.48 (0.062) | 0.59 (0.112) | 0.55 (0.055)
Statistical Analysis 1: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Natural Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.79, 95% CI 2-sided [0.45 to 0.93] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Natural Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.876, 95% CI 2-sided [0.66 to 0.96] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Natural Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.783, 95% CI 2-sided [0.17 to 0.94] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Natural Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.849, 95% CI 2-sided [-0.13 to 0.97] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Natural Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.658, 95% CI 2-sided [-0.06 to 0.93] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Natural Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.398, 95% CI 2-sided [-0.05 to 0.82] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Natural Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.776, 95% CI 2-sided [-0.02 to 0.95] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 8: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Natural Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.681, 95% CI 2-sided [-0.06 to 0.93] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 9: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Natural Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.41, 95% CI 2-sided [-0.05 to 0.83] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 10: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Fast Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.044, 95% CI 2-sided [-0.48 to 0.56] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Fast Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.938, 95% CI 2-sided [0.82 to 0.98] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Fast Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.861, 95% CI 2-sided [0.58 to 0.96] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Fast Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.392, 95% CI 2-sided [-0.14 to 0.83] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 14: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Fast Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.568, 95% CI 2-sided [-0.05 to 0.90] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 15: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Fast Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.284, 95% CI 2-sided [-0.03 to 0.74] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 16: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Fast Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.199, 95% CI 2-sided [-0.07 to 0.56] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 17: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Fast Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.657, 95% CI 2-sided [-0.04 to 0.93] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 18: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Fast Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.409, 95% CI 2-sided [-0.04 to 0.83] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 19: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Slow Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.733, 95% CI 2-sided [-0.18 to 0.94] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 20: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Slow Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.594, 95% CI 2-sided [-0.21 to 0.89] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 21: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Slow Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.392, 95% CI 2-sided [-0.21 to 0.79] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 22: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Slow Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.903, 95% CI 2-sided [0.71 to 0.97] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 23: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Slow Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.862, 95% CI 2-sided [0.62 to 0.95] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 24: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Slow Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.694, 95% CI 2-sided [0.26 to 0.90] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 25: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Slow Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.786, 95% CI 2-sided [-0.07 to 0.95] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 26: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Slow Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.694, 95% CI 2-sided [0.02 to 0.91] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 27: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Slow Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.505, 95% CI 2-sided [-0.06 to 0.83] — [estimate comment as in outcome 1, analysis 7]

4. Primary Outcome: Cohort A: Stance Duration Measured by APDM, GAITRite Walkway and ActiGraph Devices for Walk at Natural, Slow and Fast Speed Tasks
Description: Stance duration was defined as the duration of time the foot is in contact with the ground in a step during gait. Participants had to walk on GAITRite walkway (20 feet*3) wearing ActiGraph and APDM devices at participant's natural speed and at varied speeds. Natural speed was participant's self-chosen pace for 3 rounds. Varied speeds included participant's self-chosen slow pace ("Walk slow") and fast pace ("Walk fast") for 3 rounds. Raw accelerometry data collected by ActiGraph devices (comparator) was processed by the GaitPy algorithm to generate gait quality metrics (lumbar position). Gait metrics data was directly extracted from GAITRite walkway and APDM sensors (reference).
Time Frame: Up to 20 minutes on Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Cohort A: Participants Aged 3-5 Years | Cohort A: Participants Aged 6-11 Years | Cohort A: Participants Aged 12-17 Years
Number analyzed (Participants) | 13 | 14 | 13
Seconds
  ActiGraph: Natural Speed | 0.63 (0.085) | 0.65 (0.072) | 0.72 (0.054)
  GAITRite: Natural Speed | 0.64 (0.129) | 0.64 (0.082) | 0.72 (0.062)
  APDM: Natural Speed | 0.60 (0.119) | 0.59 (0.070) | 0.66 (0.065)
  ActiGraph: Fast Speed | 0.56 (0.063) | 0.58 (0.075) | 0.65 (0.046)
  GAITRite: Fast Speed | 0.49 (0.070) | 0.55 (0.087) | 0.62 (0.057)
  APDM: Fast Speed: number analyzed (Participants) | 11 | 14 | 13
  APDM: Fast Speed | 0.52 (0.050) | 0.50 (0.075) | 0.56 (0.056)
  ActiGraph: Slow Speed | 0.75 (0.081) | 0.91 (0.127) | 0.83 (0.166)
  GAITRite: Slow Speed | 0.88 (0.207) | 1.11 (0.265) | 1.02 (0.178)
  APDM: Slow Speed | 0.84 (0.205) | 1.00 (0.227) | 0.94 (0.181)
Statistical Analysis 1: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Natural Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.902, 95% CI 2-sided [0.71 to 0.97] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Natural Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.969, 95% CI 2-sided [0.90 to 0.99] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Natural Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.963, 95% CI 2-sided [0.88 to 0.99] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Natural Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.892, 95% CI 2-sided [0.58 to 0.97] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Natural Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.731, 95% CI 2-sided [-0.02 to 0.95] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Natural Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.637, 95% CI 2-sided [-0.04 to 0.92] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Natural Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.77, 95% CI 2-sided [0.36 to 0.93] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 8: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Natural Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.715, 95% CI 2-sided [-0.08 to 0.94] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 9: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Natural Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.767, 95% CI 2-sided [0.04 to 0.96] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 10: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Fast Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.24, 95% CI 2-sided [-0.18 to 0.66] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Fast Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.66, 95% CI 2-sided [-0.21 to 0.83] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Fast Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.31, 95% CI 2-sided [-0.19 to 0.72] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Fast Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.096, 95% CI 2-sided [-0.07 to 0.46] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 14: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Fast Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.1, 95% CI 2-sided [-0.01 to 0.44] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 15: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Fast Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.058, 95% CI 2-sided [-0.02 to 0.35] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 16: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Fast Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.206, 95% CI 2-sided [-0.08 to 0.59] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 17: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Fast Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.247, 95% CI 2-sided [-0.05 to 0.70] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 18: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Fast Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.127, 95% CI 2-sided [-0.03 to 0.53] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 19: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Slow Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.377, 95% CI 2-sided [-0.15 to 0.75] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 20: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Slow Speed: ActiGraph vs GAITRite; Test type: Other; Intra-class correlation coefficient = 0.44, 95% CI 2-sided [-0.21 to 0.81] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 21: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Slow Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.08, 95% CI 2-sided [-0.23 to 0.50] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 22: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Slow Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.398, 95% CI 2-sided [-0.12 to 0.76] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 23: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Slow Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.651, 95% CI 2-sided [0.04 to 0.89] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 24: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Slow Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.13, 95% CI 2-sided [-0.34 to 0.59] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 25: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Slow Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.639, 95% CI 2-sided [0.25 to 0.87] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 26: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Slow Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.666, 95% CI 2-sided [0.01 to 0.90] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 27: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Slow Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.346, 95% CI 2-sided [0.00 to 0.69] — [estimate comment as in outcome 1, analysis 7]

5. Primary Outcome: Cohort A: Swing Duration Measured by APDM, GAITRite Walkway and ActiGraph Devices for Walk at Natural, Slow and Fast Speed Tasks
Description: Swing time was defined as the time during which the foot was not in contact with the ground. Participants had to walk on GAITRite walkway (20 feet*3) wearing ActiGraph and APDM devices at participant's natural speed and at varied speeds. Natural speed was participant's self-chosen pace for 3 rounds. Varied speeds included participant's self-chosen slow pace ("Walk slow") and fast pace ("Walk fast") for 3 rounds. Raw accelerometry data collected by ActiGraph devices (comparator) was processed by the GaitPy algorithm to generate gait quality metrics (lumbar position). Gait metrics data was directly extracted from GAITRite walkway and APDM sensors (reference).
Time Frame: Up to 20 minutes on Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Cohort A: Participants Aged 3-5 Years | Cohort A: Participants Aged 6-11 Years | Cohort A: Participants Aged 12-17 Years
Number analyzed (Participants) | 13 | 14 | 13
Seconds
  Swing Duration Measured by Actigraph for Walk at Natural Speed | 0.36 (0.054) | 0.38 (0.050) | 0.42 (0.028)
  Swing Duration Measured by GAITRite for Walk at Natural Speed | 0.35 (0.034) | 0.37 (0.037) | 0.40 (0.027)
  Swing Duration Measured by APDM for Walk at Natural Speed | 0.39 (0.047) | 0.42 (0.041) | 0.45 (0.021)
  Swing Duration Measured by Actigraph for Walk at Fast Speed | 0.31 (0.030) | 0.33 (0.043) | 0.37 (0.027)
  Swing Duration Measured by GAITRite for Walk at Fast Speed | 0.30 (0.029) | 0.34 (0.039) | 0.38 (0.028)
  Swing Duration Measured by APDM for Walk at Fast Speed: number analyzed (Participants) | 11 | 14 | 13
  Swing Duration Measured by APDM for Walk at Fast Speed | 0.35 (0.025) | 0.39 (0.042) | 0.42 (0.025)
  Swing Duration Measured by Actigraph for Walk at Slow Speed: number analyzed (Participants) | 13 | 13 | 13
  Swing Duration Measured by Actigraph for Walk at Slow Speed | 0.45 (0.067) | 0.53 (0.096) | 0.56 (0.106)
  Swing Duration Measured by GAITRite for Walk at Slow Speed | 0.43 (0.058) | 0.50 (0.074) | 0.48 (0.045)
  Swing Duration Measured by APDM for Walk at Slow Speed | 0.47 (0.063) | 0.60 (0.116) | 0.55 (0.056)
Statistical Analysis 1: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Natural Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.827, 95% CI 2-sided [0.53 to 0.94] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Natural Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.877, 95% CI 2-sided [0.66 to 0.96] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Natural Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.783, 95% CI 2-sided [0.17 to 0.94] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Natural Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.833, 95% CI 2-sided [-0.14 to 0.97] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Natural Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.644, 95% CI 2-sided [-0.05 to 0.92] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Natural Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.383, 95% CI 2-sided [-0.06 to 0.81] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Natural Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.785, 95% CI 2-sided [-0.02 to 0.95] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 8: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Natural Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.679, 95% CI 2-sided [-0.06 to 0.93] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 9: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Natural Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.405, 95% CI 2-sided [-0.05 to 0.83] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 10: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Fast Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.257, 95% CI 2-sided [-0.32 to 0.69] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Fast Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.892, 95% CI 2-sided [0.69 to 0.96] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Fast Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.837, 95% CI 2-sided [0.47 to 0.95] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Fast Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.341, 95% CI 2-sided [-0.13 to 0.80] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 14: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Fast Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.536, 95% CI 2-sided [-0.05 to 0.88] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 15: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Fast Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.264, 95% CI 2-sided [-0.03 to 0.71] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 16: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Fast Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.275, 95% CI 2-sided [-0.08 to 0.66] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 17: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Fast Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.631, 95% CI 2-sided [-0.05 to 0.92] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 18: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Fast Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.379, 95% CI 2-sided [-0.03 to 0.81] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 19: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Slow Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.606, 95% CI 2-sided [0.11 to 0.86] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 20: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Slow Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.714, 95% CI 2-sided [0.29 to 0.90] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 21: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Slow Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.39, 95% CI 2-sided [-0.20 to 0.78] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 22: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Slow Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.703, 95% CI 2-sided [0.23 to 0.90] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 23: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Slow Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.555, 95% CI 2-sided [0.00 to 0.84] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 24: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Slow Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.563, 95% CI 2-sided [0.03 to 0.84] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 25: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Slow Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.687, 95% CI 2-sided [0.20 to 0.90] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 26: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Slow Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.603, 95% CI 2-sided [0.04 to 0.87] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 27: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Slow Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.459, 95% CI 2-sided [-0.02 to 0.79] — [estimate comment as in outcome 1, analysis 7]

6. Primary Outcome: Cohort A: Stride Length Measured by APDM, GAITRite Walkway and ActiGraph Devices for Walk at Natural, Slow and Fast Speed Tasks
Description: Stride length was defined as the distance covered when two steps were taken, one with each foot. It was measured from the heel of one foot to the heel of same foot when it came into contact with the ground. Participants had to walk on GAITRite walkway (20 feet*3) wearing ActiGraph and APDM devices at participant's natural speed and at varied speeds. Natural speed was participant's self-chosen pace for 3 rounds. Varied speeds included participant's self-chosen slow pace ("Walk slow") and fast pace ("Walk fast") for 3 rounds. Raw accelerometry data collected by ActiGraph devices (comparator) was processed by the GaitPy algorithm to generate gait quality metrics (lumbar position). Gait metrics data was directly extracted from GAITRite walkway and APDM sensors (reference).
Time Frame: Up to 20 minutes of Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Meters
Groups:
- Cohort A: Participants Aged 6-11 Years: Participants aged 6 to 11 years were required to wear the Actigraph centerpoint insight watch on the non-dominant wrist and lumbar region for at least 15 days. The wrist device had to be worn continuously, and the lumbar device was worn when the participants woke up in the morning and removed when they went to sleep at night or nap during the daytime. Participants also wore the APDM opal devices during Visit 1 (Day 1) only on both wrists, both feet, lumbar, and waist.
Arm/Group | Cohort A: Participants Aged 3-5 Years | Cohort A: Participants Aged 6-11 Years | Cohort A: Participants Aged 12-17 Years
Number analyzed (Participants) | 13 | 14 | 13
Meters
  ActiGraph: Natural Speed | 0.80 (0.112) | 1.01 (0.139) | 1.16 (0.146)
  GAITRite: Natural Speed | 0.89 (0.113) | 1.13 (0.127) | 1.35 (0.116)
  APDM: Natural Speed | 0.78 (0.126) | 1.02 (0.114) | 1.22 (0.118)
  ActiGraph: Fast Speed | 0.88 (0.141) | 1.12 (0.155) | 1.31 (0.109)
  GAITRite: Fast Speed | 1.02 (0.130) | 1.32 (0.195) | 1.54 (0.104)
  APDM: Fast Speed: number analyzed (Participants) | 11 | 14 | 13
  APDM: Fast Speed | 0.85 (0.144) | 1.20 (0.196) | 1.40 (0.110)
  ActiGraph: Slow Speed | 0.67 (0.122) | 0.75 (0.104) | 0.90 (0.142)
  GAITRite: Slow Speed | 0.71 (0.116) | 0.82 (0.136) | 1.08 (0.155)
  APDM: Slow Speed | 0.61 (0.118) | 0.68 (0.129) | 0.94 (0.155)
Statistical Analysis 1: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Natural Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.569, 95% CI 2-sided [-0.19 to 0.87] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Natural Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.612, 95% CI 2-sided [-0.11 to 0.91] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Natural Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.444, 95% CI 2-sided [-0.06 to 0.85] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Natural Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.254, 95% CI 2-sided [-0.35 to 0.70] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Natural Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.875, 95% CI 2-sided [0.66 to 0.96] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Natural Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.793, 95% CI 2-sided [0.02 to 0.95] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Natural Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.467, 95% CI 2-sided [0.08 to 0.78] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 8: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Natural Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.705, 95% CI 2-sided [-0.08 to 0.94] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 9: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Natural Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.585, 95% CI 2-sided [-0.05 to 0.90] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 10: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Fast Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.558, 95% CI 2-sided [-0.15 to 0.90] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Fast Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.486, 95% CI 2-sided [-0.15 to 0.87] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Fast Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.222, 95% CI 2-sided [-0.04 to 0.68] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Fast Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.729, 95% CI 2-sided [0.31 to 0.91] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 14: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Fast Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.727, 95% CI 2-sided [0.20 to 0.91] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 15: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Fast Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.592, 95% CI 2-sided [-0.19 to 0.91] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 16: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Fast Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.624, 95% CI 2-sided [-0.10 to 0.90] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 17: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Fast Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.669, 95% CI 2-sided [-0.10 to 0.92] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 18: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Fast Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.376, 95% CI 2-sided [-0.04 to 0.81] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 19: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Slow Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.755, 95% CI 2-sided [0.26 to 0.92] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 20: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Slow Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.614, 95% CI 2-sided [0.05 to 0.87] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 21: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Slow Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.424, 95% CI 2-sided [-0.18 to 0.83] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 22: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Slow Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.648, 95% CI 2-sided [0.06 to 0.89] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 23: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Slow Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.586, 95% CI 2-sided [-0.07 to 0.86] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 24: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Slow Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.759, 95% CI 2-sided [0.38 to 0.92] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 25: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Slow Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.692, 95% CI 2-sided [0.01 to 0.91] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 26: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Slow Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.614, 95% CI 2-sided [-0.08 to 0.89] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 27: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Slow Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.605, 95% CI 2-sided [-0.11 to 0.90] — [estimate comment as in outcome 1, analysis 7]

7. Primary Outcome: Cohort A: Step Duration Measured by APDM, GAITRite Walkway and ActiGraph Devices for Walk at Natural, Slow and Fast Speed Tasks
Description: Step duration was the period between the first contact of a foot and the first following contact of the contralateral foot. Participants had a single in-laboratory visit on Day 1 during which they performed gait monitoring procedures. Participants had to walk on GAITRite walkway (20 feet*3) wearing ActiGraph and APDM devices at participant's natural speed and at varied speeds. Natural speed was participant's self-chosen pace for 3 rounds. Varied speeds included participant's self-chosen slow pace ("Walk slow") and fast pace ("Walk fast") for 3 rounds. Raw accelerometry data collected by ActiGraph devices (comparator) was processed by the GaitPy algorithm to generate gait quality metrics (lumbar position). Gait metrics data was directly extracted from GAITRite walkway and APDM sensors (reference).
Time Frame: Up to 20 minutes on Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Cohort A: Participants Aged 3-5 Years | Cohort A: Participants Aged 6-11 Years | Cohort A: Participants Aged 12-17 Years
Number analyzed (Participants) | 13 | 14 | 13
Seconds
  ActiGraph: Natural Speed | 0.50 (0.072) | 0.51 (0.061) | 0.57 (0.046)
  GAITRite: Natural Speed | 0.49 (0.080) | 0.51 (0.058) | 0.56 (0.043)
  APDM: Natural Speed | 0.50 (0.081) | 0.50 (0.055) | 0.56 (0.041)
  ActiGraph: Fast Speed | 0.44 (0.061) | 0.45 (0.059) | 0.51 (0.037)
  GAITRite: Fast Speed | 0.39 (0.048) | 0.44 (0.058) | 0.50 (0.037)
  APDM: Fast Speed: number analyzed (Participants) | 11 | 14 | 13
  APDM: Fast Speed | 0.43 (0.035) | 0.44 (0.058) | 0.50 (0.038)
  ActiGraph: Slow Speed | 0.62 (0.088) | 0.76 (0.142) | 0.74 (0.109)
  GAITRite: Slow Speed | 0.65 (0.128) | 0.80 (0.163) | 0.75 (0.116)
  APDM: Slow Speed | 0.66 (0.137) | 0.80 (0.165) | 0.74 (0.116)
Statistical Analysis 1: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Natural Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.985, 95% CI 2-sided [0.94 to 1.00] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Natural Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.976, 95% CI 2-sided [0.72 to 0.99] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Natural Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.973, 95% CI 2-sided [-0.01 to 1.00] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Natural Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.984, 95% CI 2-sided [0.95 to 0.99] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Natural Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.963, 95% CI 2-sided [0.75 to 0.99] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Natural Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.945, 95% CI 2-sided [-0.16 to 0.99] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Natural Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.985, 95% CI 2-sided [0.96 to 0.99] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 8: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Natural Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.974, 95% CI 2-sided [0.91 to 0.99] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 9: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Natural Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.968, 95% CI 2-sided [0.47 to 0.99] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 10: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Fast Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = -0.019, 95% CI 2-sided [-0.39 to 0.45] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Fast Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.977, 95% CI 2-sided [-0.07 to 1.00] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Fast Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.886, 95% CI 2-sided [-0.21 to 0.98] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Fast Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.781, 95% CI 2-sided [0.42 to 0.93] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 14: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Fast Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.962, 95% CI 2-sided [0.48 to 0.99] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 15: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Fast Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.902, 95% CI 2-sided [-0.20 to 0.98] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 16: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Fast Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.21, 95% CI 2-sided [-0.07 to 0.58] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 17: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Fast Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.978, 95% CI 2-sided [0.80 to 0.99] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 18: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Fast Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.92, 95% CI 2-sided [0.12 to 0.98] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 19: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Slow Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.855, 95% CI 2-sided [0.58 to 0.95] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 20: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Slow Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.886, 95% CI 2-sided [0.52 to 0.97] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 21: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Slow Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.98, 95% CI 2-sided [0.94 to 0.99] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 22: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Slow Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.801, 95% CI 2-sided [0.42 to 0.94] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 23: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Slow Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.878, 95% CI 2-sided [0.53 to 0.96] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 24: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Slow Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.983, 95% CI 2-sided [0.94 to 0.99] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 25: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Slow Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.891, 95% CI 2-sided [0.73 to 0.96] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 26: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Slow Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.923, 95% CI 2-sided [0.77 to 0.98] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 27: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Slow Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.987, 95% CI 2-sided [0.97 to 1.00] — [estimate comment as in outcome 1, analysis 7]

8. Primary Outcome: Cohort A: Cadence Measured by APDM, GAITRite Walkway and ActiGraph Devices for Walk at Natural, Slow and Fast Speed Tasks
Description: Cadence referred to the number of steps taken per minute during gait cycle. Participants had to walk on GAITRite walkway (20 feet*3) wearing ActiGraph and APDM devices at participant's natural speed and at varied speeds. Natural speed was participant's self-chosen pace for 3 rounds. Varied speeds included participant's self-chosen slow pace ("Walk slow") and fast pace ("Walk fast") for 3 rounds. Raw accelerometry data collected by ActiGraph devices (comparator) was processed by the GaitPy algorithm to generate gait quality metrics (lumbar position). Gait metrics data was directly extracted from GAITRite walkway and APDM sensors (reference).
Time Frame: Up to 20 minutes on Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Steps per minute
Arm/Group | Cohort A: Participants Aged 3-5 Years | Cohort A: Participants Aged 6-11 Years | Cohort A: Participants Aged 12-17 Years
Number analyzed (Participants) | 13 | 14 | 13
Steps per minute
  ActiGraph: Natural Speed | 123.07 (17.515) | 118.17 (13.763) | 106.00 (7.971)
  GAITRite: Natural Speed | 120.57 (17.555) | 117.97 (14.652) | 104.23 (9.496)
  APDM: Natural Speed | 124.09 (20.093) | 120.04 (13.073) | 107.97 (7.556)
  ActiGraph: Fast Speed | 139.59 (17.740) | 134.16 (17.301) | 118.24 (8.667)
  GAITRite: Fast Speed | 147.26 (19.313) | 130.42 (16.612) | 113.16 (9.725)
  APDM: Fast Speed: number analyzed (Participants) | 11 | 14 | 13
  APDM: Fast Speed | 139.50 (10.993) | 137.06 (17.574) | 122.30 (9.326)
  ActiGraph: Slow Speed | 98.12 (14.187) | 81.48 (16.704) | 82.59 (11.866)
  GAITRite: Slow Speed | 91.77 (16.656) | 76.61 (17.346) | 81.53 (11.926)
  APDM: Slow Speed | 94.57 (17.679) | 78.38 (18.100) | 82.55 (12.486)
Statistical Analysis 1: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Natural Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.976, 95% CI 2-sided [0.74 to 0.99] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Natural Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.972, 95% CI 2-sided [0.92 to 0.99] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Natural Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.899, 95% CI 2-sided [0.66 to 0.97] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Natural Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.975, 95% CI 2-sided [0.92 to 0.99] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Natural Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.974, 95% CI 2-sided [0.80 to 0.99] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Natural Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.952, 95% CI 2-sided [-0.19 to 0.99] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Natural Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.969, 95% CI 2-sided [0.89 to 0.99] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 8: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Natural Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.968, 95% CI 2-sided [0.91 to 0.99] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 9: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Natural Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.893, 95% CI 2-sided [0.50 to 0.97] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 10: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Fast Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = -0.15, 95% CI 2-sided [-0.64 to 0.42] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Fast Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.891, 95% CI 2-sided [0.64 to 0.97] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Fast Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.561, 95% CI 2-sided [0.00 to 0.85] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Fast Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.81, 95% CI 2-sided [0.49 to 0.94] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 14: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Fast Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.967, 95% CI 2-sided [0.68 to 0.99] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 15: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Fast Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.885, 95% CI 2-sided [-0.11 to 0.98] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 16: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Fast Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.134, 95% CI 2-sided [-0.17 to 0.53] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 17: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Fast Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.896, 95% CI 2-sided [0.65 to 0.97] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 18: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Fast Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.598, 95% CI 2-sided [0.04 to 0.87] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 19: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Slow Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.849, 95% CI 2-sided [-0.09 to 0.97] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 20: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Slow Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.907, 95% CI 2-sided [0.34 to 0.98] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 21: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Slow Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.98, 95% CI 2-sided [0.92 to 0.99] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 22: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Slow Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.922, 95% CI 2-sided [0.63 to 0.98] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 23: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Slow Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.939, 95% CI 2-sided [0.76 to 0.98] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 24: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Slow Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.988, 95% CI 2-sided [0.96 to 1.00] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 25: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Slow Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.911, 95% CI 2-sided [0.61 to 0.98] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 26: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Slow Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.942, 95% CI 2-sided [0.79 to 0.98] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 27: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Slow Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.987, 95% CI 2-sided [0.96 to 1.00] — [estimate comment as in outcome 1, analysis 7]

9. Primary Outcome: Cohort A: Stride Duration Measured by APDM, GAITRite Walkway and ActiGraph Devices for Walk at Natural, Slow and Fast Speed Tasks
Description: Stride duration refers to the duration between successive heel contacts of the same foot. Participants had to walk on GAITRite walkway (20 feet*3) wearing ActiGraph and APDM devices at participant's natural speed and at varied speeds. Natural speed was participant's self-chosen pace for 3 rounds. Varied speeds included participant's self-chosen slow pace ("Walk slow") and fast pace ("Walk fast") for 3 rounds. Raw accelerometry data collected by ActiGraph devices (comparator) was processed by the GaitPy algorithm to generate gait quality metrics (lumbar position). Gait metrics data was directly extracted from GAITRite walkway and APDM sensors (reference).
Time Frame: Up to 20 minutes on Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Cohort A: Participants Aged 3-5 Years | Cohort A: Participants Aged 6-11 Years | Cohort A: Participants Aged 12-17 Years
Number analyzed (Participants) | 13 | 14 | 13
Seconds
  ActiGraph: Natural Speed | 0.99 (0.150) | 1.02 (0.118) | 1.13 (0.082)
  GAITRite: Natural Speed | 0.99 (0.162) | 1.01 (0.118) | 1.12 (0.091)
  APDM: Natural Speed | 0.99 (0.163) | 1.01 (0.111) | 1.12 (0.084)
  ActiGraph: Fast Speed | 0.88 (0.132) | 0.91 (0.115) | 1.01 (0.073)
  GAITRite: Fast Speed | 0.78 (0.093) | 0.89 (0.123) | 0.99 (0.079)
  APDM: Fast Speed: number analyzed (Participants) | 11 | 14 | 13
  APDM: Fast Speed | 0.87 (0.070) | 0.89 (0.113) | 0.99 (0.076)
  ActiGraph: Slow Speed: number analyzed (Participants) | 13 | 13 | 13
  ActiGraph: Slow Speed | 1.22 (0.155) | 1.39 (0.210) | 1.41 (0.149)
  GAITRite: Slow Speed | 1.30 (0.258) | 1.61 (0.327) | 1.49 (0.226)
  APDM: Slow Speed | 1.31 (0.265) | 1.60 (0.331) | 1.49 (0.233)
Statistical Analysis 1: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Natural Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.985, 95% CI 2-sided [0.95 to 1.00] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Natural Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.995, 95% CI 2-sided [0.09 to 1.00] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Natural Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.989, 95% CI 2-sided [0.96 to 1.00] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Natural Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.983, 95% CI 2-sided [0.95 to 0.99] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Natural Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.989, 95% CI 2-sided [0.90 to 1.00] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Natural Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.982, 95% CI 2-sided [0.28 to 1.00] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Natural Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.984, 95% CI 2-sided [0.96 to 0.99] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 8: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Natural Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.992, 95% CI 2-sided [0.97 to 1.00] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 9: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Natural Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.987, 95% CI 2-sided [0.94 to 1.00] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 10: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Fast Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = -0.092, 95% CI 2-sided [-0.44 to 0.39] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Fast Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.971, 95% CI 2-sided [0.53 to 0.99] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Fast Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.972, 95% CI 2-sided [-0.06 to 1.00] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Fast Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.725, 95% CI 2-sided [0.30 to 0.91] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 14: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Fast Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.946, 95% CI 2-sided [0.44 to 0.99] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 15: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Fast Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.939, 95% CI 2-sided [-0.12 to 0.99] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 16: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Fast Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.152, 95% CI 2-sided [-0.11 to 0.52] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 17: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Fast Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.967, 95% CI 2-sided [0.84 to 0.99] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 18: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Fast Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.965, 95% CI 2-sided [-0.04 to 0.99] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 19: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Slow Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.709, 95% CI 2-sided [0.26 to 0.90] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 20: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Slow Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.48, 95% CI 2-sided [-0.07 to 0.80] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 21: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Slow Speed: ActiGraph vs GAITRite; Test type: Other; Intraclass correlation coefficient = 0.655, 95% CI 2-sided [0.15 to 0.88] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 22: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Slow Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.692, 95% CI 2-sided [0.18 to 0.90] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 23: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Slow Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.494, 95% CI 2-sided [-0.05 to 0.81] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 24: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Slow Speed: ActiGraph vs APDM; Test type: Other; Intraclass correlation coefficient = 0.648, 95% CI 2-sided [0.16 to 0.88] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 25: Comparison: Cohort A: Participants Aged 3-5 Years; Walk at Slow Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.82, 95% CI 2-sided [0.57 to 0.94] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 26: Comparison: Cohort A: Participants Aged 6-11 Years; Walk at Slow Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.689, 95% CI 2-sided [0.30 to 0.89] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 27: Comparison: Cohort A: Participants Aged 12-17 Years; Walk at Slow Speed: ActiGraph vs GAITRite vs APDM; Test type: Other; Intraclass correlation coefficient = 0.79, 95% CI 2-sided [0.53 to 0.93] — [estimate comment as in outcome 1, analysis 7]

10. Primary Outcome: Cohort A: Double Support Duration Measured by APDM and ActiGraph Lumbar for In-lab Simulated Activities
Description: Double support time referred to the phase during walking when both feet were in contact with the ground. Participants had a single in-laboratory visit during which they performed gait monitoring procedures. For in-laboratory simulated activities, participants were required to alternate between activity blocks through a random path created by dice roll while wearing devices. Activities were done for approximately 20 minutes (approximately 7 minutes of activities [activity block 1], approximately 5 minutes of break and approximately 7 minutes of activities [activity block 2]). Activities: 2 sitting (e.g., look through a book, draw/write), 2 standing (e.g., turn a switch or hang a coat), 2 walking (e.g., move blocks/objects, toss a beanbag and pick it up). Raw accelerometry data collected by ActiGraph devices (comparator) was processed by the GaitPy algorithm to generate gait quality metrics (lumbar position). Gait metrics data was directly extracted from APDM sensors (reference).
Time Frame: Up to 20 minutes on Day 1
Population: FAS included all participants who had a signed and dated informed consent document, had assented to the study and were enrolled in the study. The outcome measure was planned to be evaluated only for Cohort A.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Cohort A: Participants Aged 3-5 Years | Cohort A: Participants Aged 6-11 Years | Cohort A: Participants Aged 12-17 Years
Number analyzed (Participants) | 13 | 14 | 13
Seconds
  APDM: Activity Block 1 | 0.22 (0.029) | 0.21 (0.061) | 0.22 (0.046)
  ActiGraph Lumbar: Activity Block 1 | 0.25 (0.013) | 0.26 (0.022) | 0.30 (0.022)
  APDM: Activity Block 2 | 0.21 (0.034) | 0.19 (0.19) | 0.21 (0.039)
  ActiGraph Lumbar: Activity Block 2 | 0.24 (0.012) | 0.27 (0.020) | 0.30 (0.023)
Statistical Analysis 1: Comparison: Cohort A: Participants Aged 3-5 Years; Activity Block 1: ActiGraph Lumbar vs APDM; Test type: Other; Intraclass correlation coefficient = 0.03, 95% CI 2-sided [-0.20 to 0.40] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohort A: Participants Aged 6-11 Years; Activity Block 1: ActiGraph Lumbar vs APDM; Test type: Other; Intraclass correlation coefficient = 0.096, 95% CI 2-sided [-0.22 to 0.50] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohort A: Participants Aged 12-17 Years; Activity Block 1: ActiGraph Lumbar vs APDM; Test type: Other; Intraclass correlation coefficient = 0.188, 95% CI 2-sided [-0.05 to 0.64] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Cohort A: Participants Aged 3-5 Years; Activity Block 2: ActiGraph Lumbar vs APDM; Test type: Other; Intraclass correlation coefficient = 0.026, 95% CI 2-sided [-0.18 to 0.39] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Cohort A: Participants Aged 6-11 Years; Activity Block 2: ActiGraph Lumbar vs APDM; Test type: Other; Intraclass correlation coefficient = 0.049, 95% CI 2-sided [-0.07 to 0.30] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Cohort A: Participants Aged 12-17 Years; Activity Block 2: ActiGraph Lumbar vs APDM; Test type: Other; Intraclass correlation coefficient = 0.144, 95% CI 2-sided [-0.04 to 0.57] — [estimate comment as in outcome 1, analysis 1]

11. Primary Outcome: Cohort A: Single Limb Support Duration Measured by APDM and ActiGraph Lumbar for In-lab Simulated Activities
Description: Single support time referred to the time when only one limb was in contact with the ground. Participants had a single in-laboratory visit during which they performed gait monitoring procedures. For in-laboratory simulated activities, participants were required to alternate between activity blocks through a random path created by dice roll while wearing devices. Activities were done for approximately 20 minutes (approximately 7 minutes of activities [activity block 1], approximately 5 minutes of break and approximately 7 minutes of activities [activity block 2]). Activities: 2 sitting (e.g., look through a book, draw/write), 2 standing (e.g., turn a switch or hang a coat), 2 walking (e.g., move blocks/objects, toss a beanbag and pick it up). Raw accelerometry data collected by ActiGraph devices (comparator) was processed by the GaitPy algorithm to generate gait quality metrics (lumbar position). Gait metrics data was directly extracted from APDM sensors (reference).
Time Frame: Up to 20 minutes on Day 1
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Cohort A: Participants Aged 3-5 Years | Cohort A: Participants Aged 6-11 Years | Cohort A: Participants Aged 12-17 Years
Number analyzed (Participants) | 13 | 14 | 13
Seconds
  APDM: Activity Block 1 | 0.37 (0.024) | 0.41 (0.038) | 0.45 (0.021)
  ActiGraph Lumbar: Activity Block 1 | 0.34 (0.017) | 0.36 (0.031) | 0.40 (0.022)
  APDM: Activity Block 2 | 0.36 (0.015) | 0.41 (0.028) | 0.44 (0.017)
  ActiGraph Lumbar: Activity Block 2 | 0.34 (0.020) | 0.36 (0.032) | 0.40 (0.024)
Statistical Analysis 1: Comparison: Cohort A: Participants Aged 3-5 Years; Activity Block 1: ActiGraph Lumbar vs APDM; Test type: Other; Intraclass correlation coefficient = 0.123, 95% CI 2-sided [-0.16 to 0.51] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohort A: Participants Aged 6-11 Years; Activity Block 1: ActiGraph Lumbar vs APDM; Test type: Other; Intraclass correlation coefficient = 0.473, 95% CI 2-sided [-0.04 to 0.86] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohort A: Participants Aged 12-17 Years; Activity Block 1: ActiGraph Lumbar vs APDM; Test type: Other; Intraclass correlation coefficient = 0.293, 95% CI 2-sided [-0.03 to 0.74] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Cohort A: Participants Aged 3-5 Years; Activity Block 2: ActiGraph Lumbar vs APDM; Test type: Other; Intraclass correlation coefficient = 0.277, 95% CI 2-sided [-0.15 to 0.73] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Cohort A: Participants Aged 6-11 Years; Activity Block 2: ActiGraph Lumbar vs APDM; Test type: Other; Intraclass correlation coefficient = 0.377, 95% CI 2-sided [-0.04 to 0.80] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Cohort A: Participants Aged 12-17 Years; Activity Block 2: ActiGraph Lumbar vs APDM; Test type: Other; Intraclass correlation coefficient = 0.279, 95% CI 2-sided [-0.03 to 0.73] — [estimate comment as in outcome 1, analysis 1]

12. Primary Outcome: Cohort A: Stance Duration Measured by APDM and ActiGraph Lumbar for In-lab Simulated Activities
Description: Stance duration was defined as the duration of time the foot is in contact with the ground in a step during gait. Participants had a single in-lab visit during which they performed gait monitoring procedures. For in-laboratory simulated activities, participants were required to alternate between activity blocks through a random path created by dice roll while wearing devices. Activities were done for approximately 20 minutes (approximately 7 minutes of activities [activity block 1], approximately 5 minutes of break and approximately 7 minutes of activities [activity block 2]). Activities: 2 sitting (e.g., look through a book, draw/write), 2 standing (e.g., turn a switch or hang a coat), 2 walking (e.g., move blocks/objects, toss a beanbag and pick it up). Raw accelerometry data collected by ActiGraph devices (comparator) was processed by the GaitPy algorithm to generate gait quality metrics (lumbar position). Gait metrics data was directly extracted from APDM sensors (reference).
Time Frame: Up to 20 minutes on Day 1
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Cohort A: Participants Aged 3-5 Years | Cohort A: Participants Aged 6-11 Years | Cohort A: Participants Aged 12-17 Years
Number analyzed (Participants) | 13 | 14 | 13
Seconds
  APDM: Activity Block 1 | 0.59 (0.044) | 0.62 (0.072) | 0.66 (0.060)
  ActiGraph Lumbar: Activity Block 1 | 0.60 (0.022) | 0.63 (0.055) | 0.72 (0.046)
  APDM: Activity Block 2 | 0.57 (0.042) | 0.60 (0.053) | 0.65 (0.053)
  ActiGraph Lumbar: Activity Block 2 | 0.60 (0.029) | 0.63 (0.051) | 0.71 (0.041)
Statistical Analysis 1: Comparison: Cohort A: Participants Aged 3-5 Years; Activity Block 1: Actigraph Lumbar vs APDM; Test type: Other; Intraclass correlation coefficient = 0.252, 95% CI 2-sided [-0.31 to 0.69] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohort A: Participants Aged 6-11 Years; Activity Block 1: Actigraph Lumbar vs APDM; Test type: Other; Intraclass correlation coefficient = 0.704, 95% CI 2-sided [0.30 to 0.89] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohort A: Participants Aged 12-17 Years; Activity Block 1: Actigraph Lumbar vs APDM; Test type: Other; Intraclass correlation coefficient = 0.631, 95% CI 2-sided [-0.09 to 0.92] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Cohort A: Participants Aged 3-5 Years; Activity Block 2: Actigraph Lumbar vs APDM; Test type: Other; Intraclass correlation coefficient = 0.292, 95% CI 2-sided [-0.18 to 0.69] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Cohort A: Participants Aged 6-11 Years; Activity Block 2: Actigraph Lumbar vs APDM; Test type: Other; Intraclass correlation coefficient = 0.516, 95% CI 2-sided [-0.07 to 0.82] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Cohort A: Participants Aged 12-17 Years; Activity Block 2: Actigraph Lumbar vs APDM; Test type: Other; Intraclass correlation coefficient = 0.566, 95% CI 2-sided [-0.04 to 0.90] — [estimate comment as in outcome 1, analysis 1]

13. Primary Outcome: Cohort A: Swing Duration Measured by APDM and ActiGraph Lumbar for In-lab Simulated Activities
Description: Swing duration was defined as the time during which the foot was not in contact with the ground. Participants had a single in-laboratory visit during which they performed gait monitoring procedures. For in-laboratory simulated activities, participants were required to alternate between activity blocks through a random path created by dice roll while wearing devices. Activities were done for approximately 20 minutes (approximately 7 minutes of activities [activity block 1], approximately 5 minutes of break and approximately 7 minutes of activities [activity block 2]). Activities: 2 sitting (e.g., look through a book, draw/write), 2 standing (e.g., turn a switch or hang a coat), 2 walking (e.g., move blocks/objects, toss a beanbag and pick it up). Raw accelerometry data collected by ActiGraph devices (comparator) was processed by the GaitPy algorithm to generate gait quality metrics (lumbar position). Gait metrics data was directly extracted from APDM sensors (reference).
Time Frame: Up to 20 minutes on Day 1
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Cohort A: Participants Aged 3-5 Years | Cohort A: Participants Aged 6-11 Years | Cohort A: Participants Aged 12-17 Years
Number analyzed (Participants) | 13 | 14 | 13
Seconds
  APDM: Activity Block 1 | 0.36 (0.020) | 0.40 (0.036) | 0.44 (0.024)
  ActiGraph Lumbar: Activity Block 1 | 0.33 (0.017) | 0.36 (0.034) | 0.40 (0.022)
  APDM: Activity Block 2 | 0.35 (0.021) | 0.40 (0.029) | 0.43 (0.019)
  ActiGraph Lumbar: Activity Block 2 | 0.33 (0.019) | 0.36 (0.030) | 0.40 (0.020)
Statistical Analysis 1: Comparison: Cohort A: Participants Aged 3-5 Years; Activity Block 1: ActiGraph Lumbar vs APDM; Test type: Other; Intra-class correlation coefficient = 0.132, 95% CI 2-sided [-0.16 to 0.52] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohort A: Participants Aged 6-11 Years; Activity Block 1: ActiGraph Lumbar vs APDM; Test type: Other; Intra-class correlation coefficient = 0.522, 95% CI 2-sided [-0.06 to 0.88] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohort A: Participants Aged 12-17 Years; Activity Block 1: ActiGraph Lumbar vs APDM; Test type: Other; Intra-class correlation coefficient = 0.363, 95% CI 2-sided [-0.06 to 0.80] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Cohort A: Participants Aged 3-5 Years; Activity Block 2: ActiGraph Lumbar vs APDM; Test type: Other; Intraclass correlation coefficient = 0.456, 95% CI 2-sided [-0.21 to 0.84] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Cohort A: Participants Aged 6-11 Years; Activity Block 2: ActiGraph Lumbar vs APDM; Test type: Other; Intraclass correlation coefficient = 0.461, 95% CI 2-sided [-0.02 to 0.85] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Cohort A: Participants Aged 12-17 Years; Activity Block 2: ActiGraph Lumbar vs APDM; Test type: Other; Intraclass correlation coefficient = 0.292, 95% CI 2-sided [-0.06 to 0.75] — [estimate comment as in outcome 1, analysis 1]

14. Primary Outcome: Cohort A: Stride Length Measured by APDM and ActiGraph Lumbar for In-lab Simulated Activities
Description: Stride length was defined as the distance covered when two steps were taken, one with each foot. It was measured from the heel of one foot to the heel of same foot when it came into contact with the ground. For in-laboratory simulated activities, participants were required to alternate between activity blocks through a random path created by dice roll while wearing devices. Activities were done for approximately 20 minutes (approximately 7 minutes of activities [activity block 1], approximately 5 minutes of break and approximately 7 minutes of activities [activity block 2]). Activities: 2 sitting (e.g., look through a book, draw/write), 2 standing (e.g., turn a switch or hang a coat), 2 walking (e.g., move blocks/objects, toss a beanbag and pick it up). Raw accelerometry data collected by ActiGraph devices (comparator) was processed by the GaitPy algorithm to generate gait quality metrics (lumbar position). Gait metrics data was directly extracted from APDM sensors (reference).
Time Frame: Up to 20 minutes on Day 1
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Meter
Arm/Group | Cohort A: Participants Aged 3-5 Years | Cohort A: Participants Aged 6-11 Years | Cohort A: Participants Aged 12-17 Years
Number analyzed (Participants) | 13 | 14 | 13
Meter
  APDM: Activity Block 1 | 0.73 (0.090) | 0.89 (0.185) | 1.12 (0.089)
  ActiGraph Lumbar: Activity Block 1 | 0.86 (0.087) | 0.99 (0.097) | 1.05 (0.110)
  APDM: Activity Block 2 | 0.71 (0.134) | 0.93 (0.165) | 1.14 (0.084)
  ActiGraph Lumbar: Activity Block 2 | 0.86 (0.094) | 1.02 (0.096) | 1.05 (0.132)
Statistical Analysis 1: Comparison: Cohort A: Participants Aged 3-5 Years; Activity Block 1: ActiGraph Lumbar vs APDM; Test type: Other; Intraclass correlation coefficient = -0.043, 95% CI 2-sided [-0.24 to 0.31] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohort A: Participants Aged 6-11 Years; Activity Block 1: ActiGraph Lumbar vs APDM; Test type: Other; Intraclass correlation coefficient = 0.284, 95% CI 2-sided [-0.19 to 0.68] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohort A: Participants Aged 12-17 Years; Activity Block 1: ActiGraph Lumbar vs APDM; Test type: Other; Intraclass correlation coefficient = 0.332, 95% CI 2-sided [-0.17 to 0.72] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Cohort A: Participants Aged 3-5 Years; Activity Block 2: ActiGraph Lumbar vs APDM; Test type: Other; Intraclass correlation coefficient = 0.041, 95% CI 2-sided [-0.22 to 0.44] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Cohort A: Participants Aged 6-11 Years; Activity Block 2: ActiGraph Lumbar vs APDM; Test type: Other; Intraclass correlation coefficient = 0.289, 95% CI 2-sided [-0.18 to 0.68] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Cohort A: Participants Aged 12-17 Years; Activity Block 2: ActiGraph Lumbar vs APDM; Test type: Other; Intraclass correlation coefficient = 0.306, 95% CI 2-sided [-0.18 to 0.70] — [estimate comment as in outcome 1, analysis 1]

15. Primary Outcome: Cohort A: Step Duration Measured by APDM and ActiGraph Lumbar for In-lab Simulated Activities
Description: Step duration was the period between the first contact of a foot and the first following contact of the contralateral foot. Participants had a single in-lab visit during which they performed gait monitoring procedures. For in-lab simulated activities, participants were required to alternate between activity blocks through a random path created by dice roll while wearing devices. Activities were done for approximately 20 minutes (approximately 7 minutes of activities [activity block 1], approximately 5 minutes of break and approximately 7 minutes of activities [activity block 2]). Activities: 2 sitting (e.g., look through a book, draw/write), 2 standing (e.g., turn a switch or hang a coat), 2 walking (e.g., move blocks/objects, toss a beanbag and pick it up). Raw accelerometry data collected by ActiGraph devices (comparator) was processed by the GaitPy algorithm to generate gait quality metrics (lumbar position). Gait metrics data was directly extracted from APDM sensors (reference).
Time Frame: Up to 20 minutes on Day 1
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Cohort A: Participants Aged 3-5 Years | Cohort A: Participants Aged 6-11 Years | Cohort A: Participants Aged 12-17 Years
Number analyzed (Participants) | 13 | 14 | 13
Seconds
  APDM: Activity Block 1 | 0.46 (0.022) | 0.50 (0.048) | 0.55 (0.039)
  ActiGraph Lumbar: Activity Block 1 | 0.47 (0.019) | 0.49 (0.045) | 0.56 (0.036)
  APDM: Activity Block 2 | 0.45 (0.021) | 0.49 (0.038) | 0.54 (0.035)
  ActiGraph Lumbar: Activity Block 2 | 0.46 (0.024) | 0.49 (0.040) | 0.55 (0.034)
Statistical Analysis 1: Comparison: Cohort A: Participants Aged 3-5 Years; Activity Block 1: ActiGraph Lumbar vs APDM; Test type: Other; Intraclass correlation coefficient = 0.596, 95% CI 2-sided [0.08 to 0.86] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohort A: Participants Aged 6-11 Years; Activity Block 1: ActiGraph Lumbar vs APDM; Test type: Other; Intraclass correlation coefficient = 0.902, 95% CI 2-sided [0.72 to 0.97] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohort A: Participants Aged 12-17 Years; Activity Block 1: ActiGraph Lumbar vs APDM; Test type: Other; Intraclass correlation coefficient = 0.944, 95% CI 2-sided [-0.15 to 0.99] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Cohort A: Participants Aged 3-5 Years; Activity Block 2: ActiGraph Lumbar vs APDM; Test type: Other; Intraclass correlation coefficient = 0.614, 95% CI 2-sided [0.10 to 0.87] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Cohort A: Participants Aged 6-11 Years; Activity Block 2: ActiGraph Lumbar vs APDM; Test type: Other; Intraclass correlation coefficient = 0.882, 95% CI 2-sided [0.67 to 0.96] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Cohort A: Participants Aged 12-17 Years; Activity Block 2: ActiGraph Lumbar vs APDM; Test type: Other; Intraclass correlation coefficient = 0.939, 95% CI 2-sided [-0.05 to 0.99] — [estimate comment as in outcome 1, analysis 1]

16. Primary Outcome: Cohort A: Cadence Measured by APDM and ActiGraph Lumbar for In-lab Simulated Activities
Description: Cadence referred to the number of steps taken per minute during gait cycle. Participants had a single in-laboratory visit during which they performed gait monitoring procedures. For in-laboratory simulated activities, participants were required to alternate between activity blocks through a random path created by dice roll while wearing devices. Activities were done for approximately 20 minutes (approximately 7 minutes of activities [activity block 1], approximately 5 minutes of break and approximately 7 minutes of activities [activity block 2]). Activities: 2 sitting (e.g., look through a book, draw/write), 2 standing (e.g., turn a switch or hang a coat), 2 walking (e.g., move blocks/objects, toss a beanbag and pick it up). Raw accelerometry data collected by ActiGraph devices (comparator) was processed by the GaitPy algorithm to generate gait quality metrics (lumbar position). Gait metrics data was directly extracted from APDM sensors (reference).
Time Frame: Up to 20 minutes on Day 1
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Steps per minute
Arm/Group | Cohort A: Participants Aged 3-5 Years | Cohort A: Participants Aged 6-11 Years | Cohort A: Participants Aged 12-17 Years
Number analyzed (Participants) | 13 | 14 | 13
Steps per minute
  APDM: Activity Block 1 | 126.97 (7.487) | 118.54 (11.395) | 109.47 (7.972)
  ActiGraph Lumbar: Activity Block 1 | 128.71 (5.515) | 122.32 (11.001) | 108.15 (6.842)
  APDM: Activity Block 2 | 130.96 (7.346) | 120.51 (8.758) | 110.84 (7.109)
  ActiGraph Lumbar: Activity Block 2 | 129.90 (6.846) | 122.49 (9.919) | 109.63 (6.715)
Statistical Analysis 1: Comparison: Cohort A: Participants Aged 3-5 Years; Activity Block 1: ActiGraph Lumbar vs APDM; Test type: Other; Intraclass correlation coefficient = 0.487, 95% CI 2-sided [-0.06 to 0.81] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohort A: Participants Aged 6-11 Years; Activity Block 1: ActiGraph Lumbar vs APDM; Test type: Other; Intraclass correlation coefficient = 0.805, 95% CI 2-sided [0.37 to 0.94] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohort A: Participants Aged 12-17 Years; Activity Block 1: ActiGraph Lumbar vs APDM; Test type: Other; Intraclass correlation coefficient = 0.953, 95% CI 2-sided [0.73 to 0.99] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Cohort A: Participants Aged 3-5 Years; Activity Block 2: ActiGraph Lumbar vs APDM; Test type: Other; Intraclass correlation coefficient = 0.584, 95% CI 2-sided [0.06 to 0.85] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Cohort A: Participants Aged 6-11 Years; Activity Block 2: ActiGraph Lumbar vs APDM; Test type: Other; Intraclass correlation coefficient = 0.785, 95% CI 2-sided [0.45 to 0.93] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Cohort A: Participants Aged 12-17 Years; Activity Block 2: ActiGraph Lumbar vs APDM; Test type: Other; Intraclass correlation coefficient = 0.964, 95% CI 2-sided [0.63 to 0.99] — [estimate comment as in outcome 1, analysis 1]

17. Primary Outcome: Cohort A: Gait Speed Measured by APDM and ActiGraph Lumbar for In-lab Simulated Activities
Description: Gait speed was the time taken to walk a specified distance. Participants had a single in-laboratory visit during which they performed gait monitoring procedures. For in-laboratory simulated activities, participants were required to alternate between activity blocks through a random path created by dice roll while wearing devices. Activities were done for approximately 20 minutes (approximately 7 minutes of activities [activity block 1], approximately 5 minutes of break and approximately 7 minutes of activities [activity block 2]). Activities: 2 sitting (e.g., look through a book, draw/write), 2 standing (e.g., turn a switch or hang a coat), 2 walking (e.g., move blocks/objects, toss a beanbag and pick it up). Raw accelerometry data collected by ActiGraph devices (comparator) was processed by the GaitPy algorithm to generate gait quality metrics (lumbar position). Gait metrics data was directly extracted from APDM sensors (reference).
Time Frame: Up to 20 minutes on Day 1
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Meters per second
Arm/Group | Cohort A: Participants Aged 3-5 Years | Cohort A: Participants Aged 6-11 Years | Cohort A: Participants Aged 12-17 Years
Number analyzed (Participants) | 13 | 14 | 13
Meters per second
  APDM: Activity Block 1 | 0.72 (0.111) | 0.80 (0.210) | 0.97 (0.109)
  ActiGraph Lumbar: Activity Block 1 | 0.91 (0.084) | 0.98 (0.085) | 0.95 (0.104)
  APDM: Activity Block 2 | 0.73 (0.158) | 0.85 (0.161) | 0.98 (0.106)
  ActiGraph Lumbar: Activity Block 2 | 0.92 (0.097) | 1.03 (0.090) | 0.96 (0.130)
Statistical Analysis 1: Comparison: Cohort A: Participants Aged 3-5 Years; Activity Block 1: ActiGraph Lumbar vs APDM; Test type: Other; Intraclass correlation coefficient = -0.023, 95% CI 2-sided [-0.16 to 0.26] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohort A: Participants Aged 6-11 Years; Activity Block 1: ActiGraph Lumbar vs APDM; Test type: Other; Intraclass correlation coefficient = 0.094, 95% CI 2-sided [-0.21 to 0.49] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohort A: Participants Aged 12-17 Years; Activity Block 1: ActiGraph Lumbar vs APDM; Test type: Other; Intraclass correlation coefficient = 0.45, 95% CI 2-sided [-0.14 to 0.80] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Cohort A: Participants Aged 3-5 Years; Activity Block 2: ActiGraph Lumbar vs APDM; Test type: Other; Intraclass correlation coefficient = -0.014, 95% CI 2-sided [-0.22 to 0.35] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Cohort A: Participants Aged 6-11 Years; Activity Block 2: ActiGraph Lumbar vs APDM; Test type: Other; Intraclass correlation coefficient = -0.13, 95% CI 2-sided [-0.35 to 0.26] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Cohort A: Participants Aged 12-17 Years; Activity Block 2: ActiGraph Lumbar vs APDM; Test type: Other; Intraclass correlation coefficient = 0.284, 95% CI 2-sided [-0.32 to 0.71] — [estimate comment as in outcome 1, analysis 1]

18. Primary Outcome: Cohort A: Total Number of Steps Measured by APDM, ActiGraph Lumbar and ActiGraph Wrist for In-lab Simulated Activities
Description: Participants had a single in-laboratory visit during which they performed gait monitoring procedures. For in-laboratory simulated activities, participants were required to alternate between activity blocks through a random path created by dice roll while wearing devices. Activities were done for approximately 20 minutes (approximately 7 minutes of activities [activity block 1], approximately 5 minutes of break and approximately 7 minutes of activities [activity block 2]). Activities: 2 sitting (e.g., look through a book, draw/write), 2 standing (e.g., turn a switch or hang a coat), 2 walking (e.g., move blocks/objects, toss a beanbag and pick it up). Raw accelerometry data collected by ActiGraph devices (comparator) was processed by the GaitPy algorithm to generate gait quality metrics (lumbar position). Gait metrics data was directly extracted from APDM sensors (reference).
Time Frame: Up to 20 minutes on Day 1
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Steps
Arm/Group | Cohort A: Participants Aged 3-5 Years | Cohort A: Participants Aged 6-11 Years | Cohort A: Participants Aged 12-17 Years
Number analyzed (Participants) | 13 | 14 | 13
Steps
  APDM: Activity Block 1 | 109.23 (42.540) | 123.00 (51.067) | 154.62 (49.399)
  ActiGraph Lumbar: Activity Block 1 | 103.00 (72.623) | 163.43 (75.572) | 114.46 (87.498)
  ActiGraph Wrist: Activity Block 1 | 187.38 (67.463) | 242.86 (73.539) | 211.15 (80.045)
  APDM: Activity Block 2 | 120.77 (57.727) | 130.57 (56.896) | 154.15 (47.430)
  ActiGraph Lumbar: Activity Block 2 | 125.46 (71.906) | 172.79 (72.707) | 109.15 (72.281)
  ActiGraph Wrist: Activity Block 2 | 210.92 (109.188) | 275.14 (87.960) | 225.69 (98.155)
Statistical Analysis 1: Comparison: Cohort A: Participants Aged 3-5 Years; Activity Block 1: ActiGraph Wrist vs APDM; Test type: Other; Intraclass correlation coefficient = 0.135, 95% CI 2-sided [-0.16 to 0.53] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohort A: Participants Aged 6-11 Years; Activity Block 1: ActiGraph Wrist vs APDM; Test type: Other; Intraclass correlation coefficient = 0.197, 95% CI 2-sided [-0.114 to 0.64] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohort A: Participants Aged 12-17 Years; Activity Block 1: ActiGraph Wrist vs APDM; Test type: Other; Intraclass correlation coefficient = 0.341, 95% CI 2-sided [-0.17 to 0.73] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Cohort A: Participants Aged 3-5 Years; Activity Block 1: ActiGraph Lumbar vs APDM; Test type: Other; Intraclass correlation coefficient = 0.38, 95% CI 2-sided [-0.23 to 0.76] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Cohort A: Participants Aged 6-11 Years; Activity Block 1: ActiGraph Lumbar vs APDM; Test type: Other; Intraclass correlation coefficient = 0.371, 95% CI 2-sided [-0.12 to 0.74] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Cohort A: Participants Aged 12-17 Years; Activity Block 1: ActiGraph Lumbar vs APDM; Test type: Other; Intraclass correlation coefficient = 0.364, 95% CI 2-sided [-0.15 to 0.74] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Cohort A: Participants Aged 3-5 Years; Activity Block 1: ActiGraph Wrist vs ActiGraph Lumbar; Test type: Other; Intraclass correlation coefficient = 0.234, 95% CI 2-sided [-0.18 to 0.65] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Cohort A: Participants Aged 6-11 Years; Activity Block 1: ActiGraph Wrist vs ActiGraph Lumbar; Test type: Other; Intraclass correlation coefficient = 0.493, 95% CI 2-sided [-0.17 to 0.87] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Cohort A: Participants Aged 12-17 Years; Activity Block 1: ActiGraph Wrist vs ActiGraph Lumbar; Test type: Other; Intraclass correlation coefficient = 0.333, 95% CI 2-sided [-0.20 to 0.75] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: Cohort A: Participants Aged 3-5 Years; Activity Block 1: ActiGraph Wrist vs ActiGraph Lumbar vs APDM; Test type: Other; Intraclass correlation coefficient = 0.228, 95% CI 2-sided [-0.06 to 0.59] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 11: Comparison: Cohort A: Participants Aged 6-11 Years; Activity Block 1: ActiGraph Wrist vs ActiGraph Lumbar vs APDM; Test type: Other; Intraclass correlation coefficient = 0.335, 95% CI 2-sided [-0.10 to 0.74] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 12: Comparison: Cohort A: Participants Aged 12-17 Years; Activity Block 1: ActiGraph Wrist vs ActiGraph Lumbar vs APDM; Test type: Other; Intraclass correlation coefficient = 0.343, 95% CI 2-sided [-0.03 to 0.70] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 13: Comparison: Cohort A: Participants Aged 3-5 Years; Activity Block 2: ActiGraph Wrist vs APDM; Test type: Other; Intraclass correlation coefficient = 0.376, 95% CI 2-sided [-0.20 to 0.77] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 14: Comparison: Cohort A: Participants Aged 6-11 Years; Activity Block 2: ActiGraph Wrist vs APDM; Test type: Other; Intraclass correlation coefficient = 0.15, 95% CI 2-sided [-0.12 to 0.56] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 15: Comparison: Cohort A: Participants Aged 12-17 Years; Activity Block 2: ActiGraph Wrist vs APDM; Test type: Other; Intraclass correlation coefficient = 0.315, 95% CI 2-sided [-0.18 to 0.71] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 16: Comparison: Cohort A: Participants Aged 3-5 Years; Activity Block 2: ActiGraph Lumbar vs APDM; Test type: Other; Intraclass correlation coefficient = 0.449, 95% CI 2-sided [-0.14 to 0.80] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 17: Comparison: Cohort A: Participants Aged 6-11 Years; Activity Block 2: ActiGraph Lumbar vs APDM; Test type: Other; Intraclass correlation coefficient = 0.241, 95% CI 2-sided [-0.22 to 0.65] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 18: Comparison: Cohort A: Participants Aged 12-17 Years; Activity Block 2: ActiGraph Lumbar vs APDM; Test type: Other; Intraclass correlation coefficient = 0.399, 95% CI 2-sided [-0.14 to 0.77] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 19: Comparison: Cohort A: Participants Aged 3-5 Years; Activity Block 2: ActiGraph Wrist vs ActiGraph Lumbar; Test type: Other; Intraclass correlation coefficient = 0.507, 95% CI 2-sided [-0.22 to 0.86] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 20: Comparison: Cohort A: Participants Aged 6-11 Years; Activity Block 2: ActiGraph Wrist vs ActiGraph Lumbar; Test type: Other; Intraclass correlation coefficient = 0.299, 95% CI 2-sided [-0.18 to 0.72] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 21: Comparison: Cohort A: Participants Aged 12-17 Years; Activity Block 2: ActiGraph Wrist vs ActiGraph Lumbar; Test type: Other; Intraclass correlation coefficient = 0.3, 95% CI 2-sided [-0.17 to 0.74] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 22: Comparison: Cohort A: Participants Aged 3-5 Years; Activity Block 2: ActiGraph Wrist vs ActiGraph Lumbar vs APDM; Test type: Other; Intraclass correlation coefficient = 0.444, 95% CI 2-sided [-0.02 to 0.78] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 23: Comparison: Cohort A: Participants Aged 6-11 Years; Activity Block 2: ActiGraph Wrist vs Actigraph Lumbar vs APDM; Test type: Other; Intraclass correlation coefficient = 0.217, 95% CI 2-sided [-0.08 to 0.59] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 24: Comparison: Cohort A: Participants Aged 12-17 Years; Activity Block 2: ActiGraph Wrist vs ActiGraph Lumbar vs APDM; Test type: Other; Intraclass correlation coefficient = 0.321, 95% CI 2-sided [-0.07 to 0.70] — [estimate comment as in outcome 1, analysis 7]

19. Primary Outcome: Cohort A: Stride Duration Measured by APDM and ActiGraph Lumbar for In-lab Simulated Activities
Description: Stride duration refers to the duration between successive heel contacts of the same foot. Participants had a single in-lab visit during which they performed gait monitoring procedures. For in-laboratory simulated activities, participants were required to alternate between activity blocks through a random path created by dice roll while wearing devices. Activities were done for approximately 20 minutes (approximately 7 minutes of activities [activity block 1], approximately 5 minutes of break and approximately 7 minutes of activities [activity block 2]). Activities: 2 sitting (e.g., look through a book, draw/write), 2 standing (e.g., turn a switch or hang a coat), 2 walking (e.g., move blocks/objects, toss a beanbag and pick it up). Raw accelerometry data collected by ActiGraph devices (comparator) was processed by the GaitPy algorithm to generate gait quality metrics (lumbar position). Gait metrics data was directly extracted from APDM sensors (reference).
Time Frame: Up to 20 minutes on Day 1
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Cohort A: Participants Aged 3-5 Years | Cohort A: Participants Aged 6-11 Years | Cohort A: Participants Aged 12-17 Years
Number analyzed (Participants) | 13 | 14 | 13
Seconds
  APDM: Activity Block 1 | 0.95 (0.060) | 1.02 (0.099) | 1.10 (0.081)
  ActiGraph Lumbar: Activity Block 1 | 0.94 (0.047) | 0.99 (0.088) | 1.10 (0.069)
  APDM: Activity Block 2 | 0.92 (0.050) | 1.00 (0.076) | 1.09 (0.070)
  ActiGraph Lumbar: Activity Block 2 | 0.93 (0.055) | 0.99 (0.079) | 1.09 (0.067)
Statistical Analysis 1: Comparison: Cohort A: Participants Aged 3-5 Years; Activity Block 1: ActiGraph Lumbar vs APDM; Test type: Other; Intraclass correlation coefficient = 0.323, 95% CI 2-sided [-0.28 to 0.73] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohort A: Participants Aged 6-11 Years; Activity Block 1: ActiGraph Lumbar vs APDM; Test type: Other; Intraclass correlation coefficient = 0.822, 95% CI 2-sided [0.23 to 0.95] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohort A: Participants Aged 12-17 Years; Activity Block 1: ActiGraph Lumbar vs APDM; Test type: Other; Intraclass correlation coefficient = 0.973, 95% CI 2-sided [0.91 to 0.99] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Cohort A: Participants Aged 3-5 Years; Activity Block 2: ActiGraph Lumbar vs APDM; Test type: Other; Intraclass correlation coefficient = 0.644, 95% CI 2-sided [0.16 to 0.88] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Cohort A: Participants Aged 6-11 Years; Activity Block 2: ActiGraph Lumbar vs APDM; Test type: Other; Intraclass correlation coefficient = 0.829, 95% CI 2-sided [0.55 to 0.94] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Cohort A: Participants Aged 12-17 Years; Activity Block 2: ActiGraph Lumbar vs APDM; Test type: Other; Intraclass correlation coefficient = 0.98, 95% CI 2-sided [0.93 to 0.99] — [estimate comment as in outcome 1, analysis 1]

20. Primary Outcome: Cohort B: Total Sleep Time During the At-Home Period
Description: Total sleep time for GeneActiv and Panoramic Bracelet was derived by the SleepPy algorithm. SleepPy algorithm was used for detecting a participant's total sleep opportunity (TSO) window and computing sleep metrics within that window.
Time Frame: From Day 1 to Day 15 (+ 3 days) for Panoramic Bracelet; Day 7 (+ 2 days) to Day 15 (+ 2 days) for GENEActiv
Population: FAS included all participants who had a signed and dated informed consent document, had assented to the study and were enrolled in the study. Here, 'Overall Number of Participants Analyzed ' signifies number of participants evaluable for this outcome measure and 'Number Analyzed' signifies number of participants analyzed for specified rows. The outcome measure was planned to be evaluated only for Cohort B.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Cohort B: Participants Aged 3-5 Years | Cohort B: Participants Aged 6-11 Years | Cohort B: Participants Aged 12-17 Years
Number analyzed (Participants) | 13 | 16 | 17
Minutes
  Panoramic Bracelet | 561.21 (43.476) | 520.34 (26.680) | 459.92 (44.421)
  GENEActiv: number analyzed (Participants) | 13 | 13 | 14
  GENEActiv | 567.48 (40.483) | 524.57 (42.583) | 450.53 (54.944)

21. Primary Outcome: Cohort B: Percentage of Time Asleep During the At-Home Period
Description: The percentage of time asleep for GeneActiv and Panoramic Bracelet was derived by the SleepPy algorithm. SleepPy algorithm was used for detecting a participant's TSO window and computing sleep metrics within that window.
Time Frame: From Day 1 to Day 15 (+ 3 days) for Panoramic Bracelet; Day 7 (+ 2 days) to Day 15 (+ 2 days) for GENEActiv
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Percentage of time
Arm/Group | Cohort B: Participants Aged 3-5 Years | Cohort B: Participants Aged 6-11 Years | Cohort B: Participants Aged 12-17 Years
Number analyzed (Participants) | 13 | 16 | 17
Percentage of time
  Panoramic Bracelet | 95.65 (1.745) | 94.93 (2.049) | 94.85 (2.481)
  GENEActiv: number analyzed (Participants) | 13 | 13 | 14
  GENEActiv | 94.85 (2.258) | 94.94 (2.402) | 94.08 (2.762)

22. Primary Outcome: Cohort B: Number of Wake Bouts During the At-Home Period
Description: Number of wake bouts for GeneActiv and Panoramic Bracelet was derived by the SleepPy algorithm. SleepPy algorithm was used for detecting a participant's TSO window and computing sleep metrics within that window.
Time Frame: From Day 1 to Day 15 (+ 3 days) for Panoramic Bracelet; Day 7 (+ 2 days) to Day 15 (+ 2 days) for GENEActiv
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Wake bouts
Arm/Group | Cohort B: Participants Aged 3-5 Years | Cohort B: Participants Aged 6-11 Years | Cohort B: Participants Aged 12-17 Years
Number analyzed (Participants) | 13 | 16 | 17
Wake bouts
  Panoramic Bracelet | 8.74 (2.895) | 9.59 (4.436) | 9.40 (4.171)
  GENEActiv: number analyzed (Participants) | 13 | 13 | 14
  GENEActiv | 9.69 (2.579) | 9.57 (4.979) | 9.37 (4.651)

23. Primary Outcome: Cohort B: Sleep Onset Latency During the At-Home Period
Description: Sleep onset latency which is time to transition from full wakefulness to sleep, for GeneActiv and Panoramic Bracelet was derived by the SleepPy algorithm. SleepPy algorithm was used for detecting a participant's TSO window and computing sleep metrics within that window.
Time Frame: From Day 1 to Day 15 (+ 3 days) for Panoramic Bracelet; Day 7 (+ 2 days) to Day 15 (+ 2 days) for GENEActiv
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Cohort B: Participants Aged 3-5 Years | Cohort B: Participants Aged 6-11 Years | Cohort B: Participants Aged 12-17 Years
Number analyzed (Participants) | 13 | 16 | 17
Minutes
  Panoramic Bracelet | 2.64 (0.868) | 3.82 (1.118) | 2.39 (1.428)
  GENEActiv: number analyzed (Participants) | 13 | 13 | 14
  GENEActiv | 3.69 (1.966) | 4.01 (1.425) | 3.64 (2.291)

24. Primary Outcome: Cohort B: Wake After Sleep Onset During the At-Home Period
Description: Wake after sleep onset is time for which participants were awake after having initially fallen asleep, for GeneActiv and Panoramic Bracelet was derived by the SleepPy algorithm. SleepPy algorithm was used for detecting a participant's TSO window and computing sleep metrics within that window.
Time Frame: From Day 1 to Day 15 (+ 3 days) for Panoramic Bracelet; Day 7 (+ 2 days) to Day 15 (+ 2 days) for GENEActiv
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Cohort B: Participants Aged 3-5 Years | Cohort B: Participants Aged 6-11 Years | Cohort B: Participants Aged 12-17 Years
Number analyzed (Participants) | 13 | 16 | 17
Minutes
  Panoramic Bracelet | 22.38 (9.022) | 24.36 (12.820) | 21.62 (12.976)
  GENEActiv: number analyzed (Participants) | 13 | 13 | 14
  GENEActiv | 26.44 (13.112) | 23.58 (15.339) | 22.01 (12.396)

25. Primary Outcome: Cohort B: Total Scratch Duration During the At-Home Period
Description: Total scratch duration for GeneActiv and Panoramic Bracelet was derived by the SleepPy algorithm. SleepPy algorithm was used for detecting a participant's TSO window and computing sleep metrics within that window.
Time Frame: From Day 1 to Day 15 (+ 3 days) for Panoramic Bracelet; Day 7 (+ 2 days) to Day 15 (+ 2 days) for GENEActiv
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Cohort B: Participants Aged 3-5 Years | Cohort B: Participants Aged 6-11 Years | Cohort B: Participants Aged 12-17 Years
Number analyzed (Participants) | 13 | 16 | 17
Minutes
  Panoramic Bracelet | 2.45 (0.785) | 3.29 (1.453) | 3.35 (1.576)
  GENEActiv: number analyzed (Participants) | 13 | 13 | 14
  GENEActiv | 3.17 (1.138) | 3.19 (1.456) | 3.75 (2.032)

26. Primary Outcome: Cohort B: Total Scratch Episodes During the At-Home Period
Description: Total scratch episodes for GeneActiv and Panoramic Bracelet was derived by the SleepPy algorithm. SleepPy algorithm was used for detecting a participant's TSO window and computing sleep metrics within that window.
Time Frame: From Day 1 to Day 15 (+ 3 days) for Panoramic Bracelet; Day 7 (+ 2 days) to Day 15 (+ 2 days) for GENEActiv
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Scratch episodes
Arm/Group | Cohort B: Participants Aged 3-5 Years | Cohort B: Participants Aged 6-11 Years | Cohort B: Participants Aged 12-17 Years
Number analyzed (Participants) | 13 | 16 | 17
Scratch episodes
  Panoramic Bracelet | 34.74 (9.585) | 45.60 (17.613) | 46.04 (19.338)
  GENEActiv: number analyzed (Participants) | 13 | 13 | 14
  GENEActiv | 43.81 (14.447) | 43.45 (16.683) | 49.74 (25.354)

27. Primary Outcome: Cohort B: Number of Available Minutes During the At-Home Period
Description: Available minutes represented any recorded accelerometer data per day per device in minutes. Number of available minutes for GENEActiv and Panoramic Bracelet was derived by the in-house built Sci-kit Digital Health (SKDH) package.
Time Frame: From Day 1 to Day 15 (+ 3 days) for Panoramic Bracelet; Day 7 (+ 2 days) to Day 15 (+ 2 days) for GENEActiv
Population: FAS included all participants who had a signed and dated informed consent document, had assented to the study and were enrolled in the study. Here, 'Number Analyzed' signifies number of participants analyzed for specified rows. The outcome measure was planned to be evaluated only for Cohort B.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Cohort B: Participants Aged 3-5 Years | Cohort B: Participants Aged 6-11 Years | Cohort B: Participants Aged 12-17 Years
Number analyzed (Participants) | 13 | 17 | 17
Minutes
  Panoramic Bracelet | 1389.08 (28.718) | 1386.44 (50.327) | 1385.76 (28.941)
  GENEActiv: number analyzed (Participants) | 13 | 13 | 14
  GENEActiv | 1234.49 (173.436) | 1260.18 (129.136) | 1310.20 (86.365)

28. Primary Outcome: Cohort B: Number of Minutes of Wear During the At-Home Period
Description: Number of minutes of wear include the total number of minutes the device is worn including sleep time and awake time. The wear time parameter (number of minutes of wear) for GENEActiv and Panoramic Bracelet was derived by the in-house built SKDH package.
Time Frame: From Day 1 to Day 15 (+ 3 days) for Panoramic Bracelet; Day 7 (+ 2 days) to Day 15 (+ 2 days) for GENEActiv
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Cohort B: Participants Aged 3-5 Years | Cohort B: Participants Aged 6-11 Years | Cohort B: Participants Aged 12-17 Years
Number analyzed (Participants) | 13 | 17 | 17
Minutes
  Panoramic Bracelet | 1095.45 (145.296) | 1099.07 (185.868) | 1044.66 (153.988)
  GENEActiv: number analyzed (Participants) | 13 | 13 | 14
  GENEActiv | 727.98 (226.617) | 785.81 (195.558) | 789.37 (181.889)

29. Primary Outcome: Cohort B: Number of Wear Minutes While Awake During the At-Home Period
Description: The wear time parameter (number of wear minutes while awake) for GENEActiv and Panoramic Bracelet was derived by the in-house built SKDH package.
Time Frame: From Day 1 to Day 15 (+ 3 days) for Panoramic Bracelet; Day 7 (+ 2 days) to Day 15 (+ 2 days) for GENEActiv
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Cohort B: Participants Aged 3-5 Years | Cohort B: Participants Aged 6-11 Years | Cohort B: Participants Aged 12-17 Years
Number analyzed (Participants) | 13 | 17 | 17
Minutes
  Panoramic Bracelet | 813.15 (47.851) | 883.23 (73.627) | 845.01 (85.179)
  GENEActiv: number analyzed (Participants) | 13 | 13 | 14
  GENEActiv | 706.48 (85.259) | 768.64 (99.152) | 775.16 (152.259)

30. Primary Outcome: Cohort B: Number of Participants According to Response to At-home Wearability/Comfort Questionnaire for Panoramic Bracelet Device at Day 7
Description: Wearability/comfort questionnaire included a total of 10 items for which the participants (12 to 17 years) or their caregivers (participants aged 3 to 11 years) were required to provide a response on a scale of 0 to 4, where 0 = strongly disagree, and 4 = strongly agree, higher scores indicated more comfort, except for questions 5 ("The device changes the way I move") and 6 ("The device changes the way I behave") , where 0 = strongly agree and 4 = strongly disagree, higher scores indicate more comfort. Number of participants according to response to each item of the wearability/comfort questionnaire is reported.
Time Frame: Day 7
Population: FAS included all participants who had a signed and dated informed consent document, had assented to the study and were enrolled in the study. The outcome measure was planned to be evaluated only for Cohort B.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort B: Participants Aged 3-5 Years | Cohort B: Participants Aged 6-11 Years | Cohort B: Participants Aged 12-17 Years
Number analyzed (Participants) | 13 | 17 | 17
Participants
  Comfortable to Wear: 0 | 0 | 0 | 0
  Comfortable to Wear: 1 | 1 | 1 | 0
  Comfortable to Wear: 2 | 1 | 1 | 1
  Comfortable to Wear: 3 | 6 | 8 | 11
  Comfortable to Wear: 4 | 5 | 7 | 5
  Easy to Put On: 0 | 0 | 0 | 0
  Easy to Put On: 1 | 0 | 1 | 1
  Easy to Put On: 2 | 0 | 3 | 2
  Easy to Put On: 3 | 9 | 7 | 7
  Easy to Put On: 4 | 4 | 6 | 7
  Easy to Take Off: 0 | 0 | 0 | 0
  Easy to Take Off: 1 | 0 | 0 | 0
  Easy to Take Off: 2 | 0 | 3 | 0
  Easy to Take Off: 3 | 7 | 7 | 7
  Easy to Take Off: 4 | 6 | 7 | 10
  Easy to Wear: 0 | 0 | 0 | 0
  Easy to Wear: 1 | 0 | 1 | 0
  Easy to Wear: 2 | 2 | 2 | 0
  Easy to Wear: 3 | 8 | 7 | 6
  Easy to Wear: 4 | 3 | 7 | 11
  Changes the Way I Move: 0 | 0 | 0 | 0
  Changes the Way I Move: 1 | 0 | 0 | 0
  Changes the Way I Move: 2 | 0 | 0 | 0
  Changes the Way I Move: 3 | 6 | 5 | 3
  Changes the Way I Move: 4 | 7 | 12 | 14
  Changes the Way I Behave: 0 | 0 | 0 | 0
  Changes the Way I Behave: 1 | 0 | 0 | 0
  Changes the Way I Behave: 2 | 0 | 0 | 0
  Changes the Way I Behave: 3 | 6 | 7 | 4
  Changes the Way I Behave: 4 | 7 | 10 | 13
  Willing to Wear for 4 to 7 Days: 0 | 0 | 0 | 0
  Willing to Wear for 4 to 7 Days: 1 | 0 | 1 | 0
  Willing to Wear for 4 to 7 Days: 2 | 0 | 0 | 0
  Willing to Wear for 4 to 7 Days: 3 | 7 | 5 | 8
  Willing to Wear for 4 to 7 Days: 4 | 6 | 11 | 9
  Willing to Wear for > 7 Days: 0 | 0 | 0 | 0
  Willing to Wear for > 7 Days: 1 | 0 | 1 | 0
  Willing to Wear for > 7 Days: 2 | 0 | 0 | 0
  Willing to Wear for > 7 Days: 3 | 9 | 8 | 9
  Willing to Wear for > 7 Days: 4 | 4 | 8 | 8
  If the device could follow my progress during a treatment (ttmt), I would wear it: 0 | 0 | 0 | 0
  If the device could follow my progress during a treatment (ttmt), I would wear it: 1 | 0 | 0 | 0
  If the device could follow my progress during a treatment (ttmt), I would wear it: 2 | 1 | 1 | 0
  If the device could follow my progress during a treatment (ttmt), I would wear it: 3 | 5 | 8 | 6
  If the device could follow my progress during a treatment (ttmt), I would wear it: 4 | 7 | 8 | 11
  If device could follow my progress during ttmt, I would want my doctor to have access to my results: 0 | 0 | 0 | 0
  If device could follow my progress during ttmt, I would want my doctor to have access to my results: 1 | 0 | 0 | 0
  If device could follow my progress during ttmt, I would want my doctor to have access to my results: 2 | 0 | 0 | 0
  If device could follow my progress during ttmt, I would want my doctor to have access to my results: 3 | 6 | 9 | 6
  If device could follow my progress during ttmt, I would want my doctor to have access to my results: 4 | 7 | 8 | 11

31. Secondary Outcome: Cohort A: Number of Participants Enrolled Over Time
Description: Number of participants enrolled at specified month intervals in the study is reported in this outcome measure.
Time Frame: Up to approximately 8 months
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Participants Aged 3-5 Years | Cohort A: Participants Aged 6-11 Years | Cohort A: Participants Aged 12-17 Years
Number analyzed (Participants) | 13 | 14 | 13
Participants
  23-Aug-2021 to 22-Sep-2021 | 5 | 3 | 5
  23-Sep-2021 to 22-Oct-2021 | 2 | 6 | 5
  23-Oct-2021 to 22-Nov-2021 | 1 | 3 | 3
  23-Nov-2021 to 22-Dec-2021 | 0 | 2 | 0
  23-Dec-2021 to 22-Jan-2022 | 1 | 0 | 0
  23-Jan-2022 to 22-Feb-2022 | 0 | 0 | 0
  23-Feb-2022 to 22-Mar-2022 | 1 | 0 | 0
  23-Mar-2022 to 22-Apr-2022 | 3 | 0 | 0

32. Primary Outcome: Cohort A: Number of Days to Complete Enrollment
Description: Number of days to complete enrollment corresponded to the total number of days it took to enroll all study participants within the age groups of 3-5 years, 6-11 years and 12-17 years.
Time Frame: Up to approximately 8 months
Population: as for outcome 10
Measure: Number; unit: Days
Arm/Group | Cohort A: Participants Aged 3-5 Years | Cohort A: Participants Aged 6-11 Years | Cohort A: Participants Aged 12-17 Years
Number analyzed (Participants) | 13 | 14 | 13
Days | 232 | 101 | 77

33. Secondary Outcome: Cohort A: Number of Participants Able to Perform Each of the 7 Lab-Based Tasks
Description: Number of participants who were able to perform each of the 7 tasks (i.e., walking at natural, slow and fast speeds, tile and carpet walks, 2 sessions of in-lab simulated activities) is reported in this outcome measure.
Time Frame: Up to 20 minutes on Day 1
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Participants Aged 3-5 Years | Cohort A: Participants Aged 6-11 Years | Cohort A: Participants Aged 12-17 Years
Number analyzed (Participants) | 13 | 14 | 13
Participants
  Natural Walk | 13 | 14 | 13
  Fast Walk | 13 | 14 | 13
  Slow Walk | 13 | 14 | 13
  Carpet Walk | 13 | 14 | 13
  Tile Walk | 13 | 14 | 13
  Activity Block 1 | 13 | 14 | 13
  Activity Block 2 | 13 | 14 | 13

34. Secondary Outcome: Cohort A: Percentage of Tasks Completed (From a Total of 7 Tasks)
Description: Percentage of tasks completed from a total of 7 tasks (i.e., walking at natural, slow and fast speeds, tile and carpet walks, 2 sessions of in-lab simulated activities) is reported in this outcome measure.
Time Frame: Up to 20 minutes on Day 1
Population: as for outcome 10
Measure: Median (Full Range); unit: Percentage of tasks
Arm/Group | Cohort A: Participants Aged 3-5 Years | Cohort A: Participants Aged 6-11 Years | Cohort A: Participants Aged 12-17 Years
Number analyzed (Participants) | 13 | 14 | 13
Percentage of tasks | 100 [100 to 100] | 100 [100 to 100] | 100 [100 to 100]

35. Secondary Outcome: Cohort A: Number of Hours Per Day Wearing the Lumbar and Wrist Devices
Time Frame: From Day 1 to Day 15 (+ 3 days)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Hours per day
Arm/Group | Cohort A: Participants Aged 3-5 Years | Cohort A: Participants Aged 6-11 Years | Cohort A: Participants Aged 12-17 Years
Number analyzed (Participants) | 13 | 14 | 13
Hours per day
  Wrist device | 21.05 (2.461) | 21.80 (1.947) | 22.01 (2.169)
  Lumbar device | 7.24 (4.293) | 12.51 (3.630) | 14.24 (4.574)

36. Secondary Outcome: Cohort A: Number of Days With More Than 10 Hours of Wear Time for Lumbar Device
Time Frame: From Day 1 to Day 15 (+ 3 days)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Cohort A: Participants Aged 3-5 Years | Cohort A: Participants Aged 6-11 Years | Cohort A: Participants Aged 12-17 Years
Number analyzed (Participants) | 13 | 14 | 13
Days | 6.15 (4.413) | 11.71 (3.561) | 11.69 (2.250)

37. Secondary Outcome: Cohort A: Number of Days With More Than 18 Hours of Wear Time for Wrist Device
Time Frame: From Day 1 to Day 15 (+ 3 days)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Cohort A: Participants Aged 3-5 Years | Cohort A: Participants Aged 6-11 Years | Cohort A: Participants Aged 12-17 Years
Number analyzed (Participants) | 13 | 14 | 13
Days | 12.38 (2.534) | 13.21 (1.718) | 12.54 (2.436)

38. Secondary Outcome: Cohort A: Number of Participants According to Response to In Lab Wearability/Comfort Questionnaire for APDM Device and for ActiGraph Lumbar and Wrist Device at Day 1
Description: Wearability/comfort questionnaire included a total of 10 items for which the participants (12 to 17 years) or their caregivers (participants aged 3 to 11 years) were required to provide a response on a scale of 0 to 4, where 0 = strongly disagree, and 4 = strongly agree, higher scores indicate more comfort except for questions 5 ("The device changes the way I move") and 6 ("The device changes the way I behave") , where 0 = strongly agree and 4 = strongly disagree, higher scores indicate more comfort. Number of participants according to response to each item of the wearability/comfort questionnaire is reported.
Time Frame: Day 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Participants Aged 3-5 Years | Cohort A: Participants Aged 6-11 Years | Cohort A: Participants Aged 12-17 Years
Number analyzed (Participants) | 13 | 14 | 13
Participants
  APDM: Comfortable to Wear: 0 | 1 | 0 | 0
  APDM: Comfortable to Wear: 1 | 0 | 0 | 1
  APDM: Comfortable to Wear: 2 | 2 | 1 | 5
  APDM: Comfortable to Wear: 3 | 4 | 9 | 6
  APDM: Comfortable to Wear: 4 | 6 | 4 | 1
  APDM: Easy to Put On: 0 | 1 | 0 | 0
  APDM: Easy to Put On: 1 | 0 | 0 | 1
  APDM: Easy to Put On: 2 | 1 | 4 | 5
  APDM: Easy to Put On: 3 | 5 | 4 | 6
  APDM: Easy to Put On: 4 | 6 | 6 | 1
  APDM: Easy to Take Off: 0 | 1 | 0 | 0
  APDM: Easy to Take Off: 1 | 0 | 0 | 3
  APDM: Easy to Take Off: 2 | 0 | 1 | 2
  APDM: Easy to Take Off: 3 | 6 | 6 | 6
  APDM: Easy to Take Off: 4 | 6 | 7 | 2
  APDM: Easy to Wear: 0 | 1 | 0 | 0
  APDM: Easy to Wear: 1 | 0 | 0 | 0
  APDM: Easy to Wear: 2 | 1 | 2 | 1
  APDM: Easy to Wear: 3 | 7 | 6 | 9
  APDM: Easy to Wear: 4 | 4 | 6 | 3
  APDM: Changes the Way I Move: 0 | 0 | 0 | 0
  APDM: Changes the Way I Move: 1 | 1 | 1 | 0
  APDM: Changes the Way I Move: 2 | 1 | 0 | 4
  APDM: Changes the Way I Move: 3 | 7 | 2 | 6
  APDM: Changes the Way I Move: 4 | 4 | 11 | 3
  APDM: Changes the Way I Behave: 0 | 0 | 0 | 0
  APDM: Changes the Way I Behave: 1 | 2 | 0 | 0
  APDM: Changes the Way I Behave: 2 | 0 | 0 | 1
  APDM: Changes the Way I Behave: 3 | 6 | 1 | 7
  APDM: Changes the Way I Behave: 4 | 5 | 13 | 5
  APDM: Willing to Wear for 4 to 7 Days: 0 | 0 | 0 | 0
  APDM: Willing to Wear for 4 to 7 Days: 1 | 3 | 0 | 1
  APDM: Willing to Wear for 4 to 7 Days: 2 | 0 | 3 | 0
  APDM: Willing to Wear for 4 to 7 Days: 3 | 6 | 4 | 9
  APDM: Willing to Wear for 4 to 7 Days: 4 | 4 | 7 | 3
  APDM: Willing to Wear for > 7 Days: 0 | 1 | 0 | 0
  APDM: Willing to Wear for > 7 Days: 1 | 2 | 1 | 1
  APDM: Willing to Wear for > 7 Days: 2 | 3 | 1 | 3
  APDM: Willing to Wear for > 7 Days: 3 | 3 | 6 | 7
  APDM: Willing to Wear for > 7 Days: 4 | 4 | 6 | 2
  APDM: If the device could follow my progress during a treatment, I would wear it: 0 | 0 | 0 | 0
  APDM: If the device could follow my progress during a treatment, I would wear it: 1 | 2 | 0 | 0
  APDM: If the device could follow my progress during a treatment, I would wear it: 2 | 0 | 0 | 0
  APDM: If the device could follow my progress during a treatment, I would wear it: 3 | 5 | 6 | 5
  APDM: If the device could follow my progress during a treatment, I would wear it: 4 | 6 | 8 | 8
  APDM: If device could follow my progress during ttmt, I want my doctor to have access to my results: 0 | 0 | 0 | 0
  APDM: If device could follow my progress during ttmt, I want my doctor to have access to my results: 1 | 0 | 0 | 0
  APDM: If device could follow my progress during ttmt, I want my doctor to have access to my results: 2 | 0 | 0 | 0
  APDM: If device could follow my progress during ttmt, I want my doctor to have access to my results: 3 | 5 | 5 | 6
  APDM: If device could follow my progress during ttmt, I want my doctor to have access to my results: 4 | 8 | 9 | 7
  ActiGraph (ACT) Lumbar (L): Comfortable to Wear: 0 | 0 | 0 | 0
  ActiGraph (ACT) Lumbar (L): Comfortable to Wear: 1 | 1 | 0 | 1
  ActiGraph (ACT) Lumbar (L): Comfortable to Wear: 2 | 0 | 1 | 3
  ActiGraph (ACT) Lumbar (L): Comfortable to Wear: 3 | 6 | 8 | 8
  ActiGraph (ACT) Lumbar (L): Comfortable to Wear: 4 | 6 | 5 | 1
  ACT L: Easy to Put On: 0 | 0 | 0 | 0
  ACT L: Easy to Put On: 1 | 1 | 0 | 0
  ACT L: Easy to Put On: 2 | 0 | 1 | 4
  ACT L: Easy to Put On: 3 | 5 | 4 | 7
  ACT L: Easy to Put On: 4 | 7 | 9 | 2
  ACT L: Easy to Take Off: 0 | 0 | 0 | 0
  ACT L: Easy to Take Off: 1 | 0 | 0 | 0
  ACT L: Easy to Take Off: 2 | 0 | 1 | 1
  ACT L: Easy to Take Off: 3 | 5 | 2 | 7
  ACT L: Easy to Take Off: 4 | 8 | 11 | 5
  ACT L: Easy to Wear: 0 | 0 | 0 | 0
  ACT L: Easy to Wear: 1 | 1 | 0 | 0
  ACT L: Easy to Wear: 2 | 0 | 0 | 1
  ACT L: Easy to Wear: 3 | 5 | 6 | 8
  ACT L: Easy to Wear: 4 | 7 | 8 | 4
  ACT L: Changes the Way I Move: 0 | 0 | 0 | 0
  ACT L: Changes the Way I Move: 1 | 0 | 0 | 0
  ACT L: Changes the Way I Move: 2 | 0 | 0 | 1
  ACT L: Changes the Way I Move: 3 | 4 | 2 | 7
  ACT L: Changes the Way I Move: 4 | 9 | 12 | 5
  ACT L: Changes the Way I Behave: 0 | 0 | 0 | 0
  ACT L: Changes the Way I Behave: 1 | 0 | 0 | 0
  ACT L: Changes the Way I Behave: 2 | 1 | 0 | 0
  ACT L: Changes the Way I Behave: 3 | 3 | 1 | 5
  ACT L: Changes the Way I Behave: 4 | 9 | 13 | 8
  ACT L: Willing to Wear for 4 to 7 Days: 0 | 0 | 0 | 0
  ACT L: Willing to Wear for 4 to 7 Days: 1 | 0 | 0 | 0
  ACT L: Willing to Wear for 4 to 7 Days: 2 | 0 | 0 | 0
  ACT L: Willing to Wear for 4 to 7 Days: 3 | 6 | 3 | 5
  ACT L: Willing to Wear for 4 to 7 Days: 4 | 7 | 11 | 8
  ACT L: Willing to Wear for > 7 Days: 0 | 0 | 0 | 0
  ACT L: Willing to Wear for > 7 Days: 1 | 0 | 0 | 0
  ACT L: Willing to Wear for > 7 Days: 2 | 0 | 0 | 2
  ACT L: Willing to Wear for > 7 Days: 3 | 7 | 4 | 3
  ACT L: Willing to Wear for > 7 Days: 4 | 6 | 10 | 8
  ACT L: If the device could follow my progress during a treatment, I would wear it: 0 | 0 | 0 | 0
  ACT L: If the device could follow my progress during a treatment, I would wear it: 1 | 0 | 0 | 0
  ACT L: If the device could follow my progress during a treatment, I would wear it: 2 | 0 | 0 | 0
  ACT L: If the device could follow my progress during a treatment, I would wear it: 3 | 6 | 4 | 5
  ACT L: If the device could follow my progress during a treatment, I would wear it: 4 | 7 | 10 | 8
  ACT L:If device could follow my progress during ttmt, I want my doctor to have access to my results: 0 | 0 | 0 | 0
  ACT L:If device could follow my progress during ttmt, I want my doctor to have access to my results: 1 | 0 | 0 | 0
  ACT L:If device could follow my progress during ttmt, I want my doctor to have access to my results: 2 | 0 | 0 | 0
  ACT L:If device could follow my progress during ttmt, I want my doctor to have access to my results: 3 | 4 | 5 | 6
  ACT L:If device could follow my progress during ttmt, I want my doctor to have access to my results: 4 | 9 | 9 | 7
  ActiGraph (ACT) Wrist (W): Comfortable to Wear: 0 | 0 | 0 | 0
  ActiGraph (ACT) Wrist (W): Comfortable to Wear: 1 | 1 | 0 | 0
  ActiGraph (ACT) Wrist (W): Comfortable to Wear: 2 | 1 | 2 | 2
  ActiGraph (ACT) Wrist (W): Comfortable to Wear: 3 | 3 | 4 | 8
  ActiGraph (ACT) Wrist (W): Comfortable to Wear: 4 | 8 | 8 | 3
  ACT W: Easy to Put On: 0 | 1 | 0 | 0
  ACT W: Easy to Put On: 1 | 1 | 0 | 1
  ACT W: Easy to Put On: 2 | 0 | 0 | 2
  ACT W: Easy to Put On: 3 | 2 | 6 | 5
  ACT W: Easy to Put On: 4 | 9 | 8 | 5
  ACT W: Easy to Take Off: 0 | 0 | 0 | 0
  ACT W: Easy to Take Off: 1 | 0 | 0 | 1
  ACT W: Easy to Take Off: 2 | 0 | 0 | 1
  ACT W: Easy to Take Off: 3 | 4 | 8 | 4
  ACT W: Easy to Take Off: 4 | 9 | 6 | 7
  ACT W: Easy to Wear: number analyzed (Participants) | 13 | 14 | 12
  ACT W: Easy to Wear: 0 | 0 | 0 | 0
  ACT W: Easy to Wear: 1 | 0 | 0 | 0
  ACT W: Easy to Wear: 2 | 0 | 1 | 0
  ACT W: Easy to Wear: 3 | 7 | 6 | 6
  ACT W: Easy to Wear: 4 | 6 | 7 | 6
  ACT W: Changes the Way I Move: 0 | 0 | 0 | 1
  ACT W: Changes the Way I Move: 1 | 0 | 0 | 0
  ACT W: Changes the Way I Move: 2 | 2 | 0 | 0
  ACT W: Changes the Way I Move: 3 | 4 | 4 | 5
  ACT W: Changes the Way I Move: 4 | 7 | 10 | 7
  ACT W: Changes the Way I Behave: 0 | 0 | 0 | 0
  ACT W: Changes the Way I Behave: 1 | 1 | 0 | 0
  ACT W: Changes the Way I Behave: 2 | 2 | 0 | 0
  ACT W: Changes the Way I Behave: 3 | 2 | 3 | 3
  ACT W: Changes the Way I Behave: 4 | 8 | 11 | 10
  ACT W: Willing to Wear for 4 to 7 Days: 0 | 0 | 0 | 0
  ACT W: Willing to Wear for 4 to 7 Days: 1 | 0 | 0 | 0
  ACT W: Willing to Wear for 4 to 7 Days: 2 | 0 | 0 | 0
  ACT W: Willing to Wear for 4 to 7 Days: 3 | 4 | 3 | 4
  ACT W: Willing to Wear for 4 to 7 Days: 4 | 9 | 11 | 9
  ACT W: Willing to Wear for > 7 Days: 0 | 0 | 0 | 0
  ACT W: Willing to Wear for > 7 Days: 1 | 0 | 0 | 0
  ACT W: Willing to Wear for > 7 Days: 2 | 1 | 0 | 0
  ACT W: Willing to Wear for > 7 Days: 3 | 7 | 3 | 4
  ACT W: Willing to Wear for > 7 Days: 4 | 5 | 11 | 9
  ACT W: If the device could follow my progress during a ttmt, I would wear it: 0 | 0 | 0 | 0
  ACT W: If the device could follow my progress during a ttmt, I would wear it: 1 | 0 | 0 | 0
  ACT W: If the device could follow my progress during a ttmt, I would wear it: 2 | 0 | 0 | 0
  ACT W: If the device could follow my progress during a ttmt, I would wear it: 3 | 5 | 3 | 4
  ACT W: If the device could follow my progress during a ttmt, I would wear it: 4 | 8 | 11 | 9
  ACT W:If device could follow my progress during ttmt, I want my doctor to have access to my results: 0 | 0 | 0 | 0
  ACT W:If device could follow my progress during ttmt, I want my doctor to have access to my results: 1 | 0 | 0 | 0
  ACT W:If device could follow my progress during ttmt, I want my doctor to have access to my results: 2 | 0 | 0 | 0
  ACT W:If device could follow my progress during ttmt, I want my doctor to have access to my results: 3 | 3 | 4 | 6
  ACT W:If device could follow my progress during ttmt, I want my doctor to have access to my results: 4 | 10 | 10 | 7

39. Secondary Outcome: Cohort A: Number of Participants According to Response to At-home Wearability/Comfort Questionnaire for ActiGraph Lumbar and Wrist Device at Final Study Evaluation
Description: as for outcome 38
Time Frame: Day 15 (+ 3 days)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Participants Aged 3-5 Years | Cohort A: Participants Aged 6-11 Years | Cohort A: Participants Aged 12-17 Years
Number analyzed (Participants) | 13 | 14 | 13
Participants
  ActiGraph (ACT) Lumbar (L): Comfortable to Wear: 0 | 1 | 0 | 0
  ActiGraph (ACT) Lumbar (L): Comfortable to Wear: 1 | 2 | 0 | 2
  ActiGraph (ACT) Lumbar (L): Comfortable to Wear: 2 | 0 | 2 | 4
  ActiGraph (ACT) Lumbar (L): Comfortable to Wear: 3 | 7 | 8 | 3
  ActiGraph (ACT) Lumbar (L): Comfortable to Wear: 4 | 3 | 4 | 4
  ACT L: Easy to Put On: 0 | 0 | 0 | 0
  ACT L: Easy to Put On: 1 | 0 | 1 | 1
  ACT L: Easy to Put On: 2 | 1 | 0 | 1
  ACT L: Easy to Put On: 3 | 5 | 5 | 3
  ACT L: Easy to Put On: 4 | 7 | 8 | 8
  ACT L: Easy to Take Off: 0 | 0 | 0 | 0
  ACT L: Easy to Take Off: 1 | 0 | 0 | 0
  ACT L: Easy to Take Off: 2 | 1 | 0 | 0
  ACT L: Easy to Take Off: 3 | 4 | 5 | 3
  ACT L: Easy to Take Off: 4 | 8 | 9 | 10
  ACT L: Easy to Wear: 0 | 0 | 0 | 0
  ACT L: Easy to Wear: 1 | 1 | 1 | 1
  ACT L: Easy to Wear: 2 | 2 | 2 | 4
  ACT L: Easy to Wear: 3 | 7 | 5 | 2
  ACT L: Easy to Wear: 4 | 3 | 6 | 6
  ACT L: Changes the Way I Move: 0 | 0 | 0 | 0
  ACT L: Changes the Way I Move: 1 | 1 | 2 | 0
  ACT L: Changes the Way I Move: 2 | 0 | 0 | 0
  ACT L: Changes the Way I Move: 3 | 6 | 3 | 6
  ACT L: Changes the Way I Move: 4 | 6 | 9 | 7
  ACT L: Changes the Way I Behave: 0 | 0 | 0 | 0
  ACT L: Changes the Way I Behave: 1 | 1 | 1 | 0
  ACT L: Changes the Way I Behave: 2 | 0 | 1 | 0
  ACT L: Changes the Way I Behave: 3 | 5 | 2 | 4
  ACT L: Changes the Way I Behave: 4 | 7 | 10 | 9
  ACT L: Willing to Wear for 4 to 7 Days: 0 | 1 | 0 | 0
  ACT L: Willing to Wear for 4 to 7 Days: 1 | 2 | 1 | 0
  ACT L: Willing to Wear for 4 to 7 Days: 2 | 0 | 0 | 0
  ACT L: Willing to Wear for 4 to 7 Days: 3 | 7 | 6 | 5
  ACT L: Willing to Wear for 4 to 7 Days: 4 | 3 | 7 | 8
  ACT L: Willing to Wear for > 7 Days: 0 | 2 | 0 | 0
  ACT L: Willing to Wear for > 7 Days: 1 | 2 | 1 | 0
  ACT L: Willing to Wear for > 7 Days: 2 | 1 | 0 | 1
  ACT L: Willing to Wear for > 7 Days: 3 | 5 | 8 | 4
  ACT L: Willing to Wear for > 7 Days: 4 | 3 | 5 | 8
  ACT L: If the device could follow my progress during a treatment, I would wear it: 0 | 0 | 0 | 0
  ACT L: If the device could follow my progress during a treatment, I would wear it: 1 | 1 | 0 | 0
  ACT L: If the device could follow my progress during a treatment, I would wear it: 2 | 0 | 0 | 0
  ACT L: If the device could follow my progress during a treatment, I would wear it: 3 | 6 | 5 | 3
  ACT L: If the device could follow my progress during a treatment, I would wear it: 4 | 6 | 9 | 10
  ACT L:If device could follow my progress during ttmt, I want my doctor to have access to my results: 0 | 0 | 0 | 0
  ACT L:If device could follow my progress during ttmt, I want my doctor to have access to my results: 1 | 0 | 0 | 0
  ACT L:If device could follow my progress during ttmt, I want my doctor to have access to my results: 2 | 0 | 0 | 0
  ACT L:If device could follow my progress during ttmt, I want my doctor to have access to my results: 3 | 3 | 4 | 4
  ACT L:If device could follow my progress during ttmt, I want my doctor to have access to my results: 4 | 10 | 10 | 9
  ActiGraph (ACT) Wrist (W): Comfortable to Wear: 0 | 0 | 0 | 0
  ActiGraph (ACT) Wrist (W): Comfortable to Wear: 1 | 1 | 0 | 0
  ActiGraph (ACT) Wrist (W): Comfortable to Wear: 2 | 0 | 0 | 1
  ActiGraph (ACT) Wrist (W): Comfortable to Wear: 3 | 5 | 5 | 5
  ActiGraph (ACT) Wrist (W): Comfortable to Wear: 4 | 7 | 9 | 7
  ACT W: Easy to Put On: 0 | 0 | 0 | 0
  ACT W: Easy to Put On: 1 | 1 | 1 | 0
  ACT W: Easy to Put On: 2 | 0 | 1 | 1
  ACT W: Easy to Put On: 3 | 4 | 6 | 5
  ACT W: Easy to Put On: 4 | 8 | 6 | 7
  ACT W: Easy to Take Off: 0 | 0 | 0 | 0
  ACT W: Easy to Take Off: 1 | 1 | 0 | 0
  ACT W: Easy to Take Off: 2 | 0 | 0 | 0
  ACT W: Easy to Take Off: 3 | 4 | 8 | 4
  ACT W: Easy to Take Off: 4 | 8 | 6 | 9
  ACT W: Easy to Wear: 0 | 0 | 0 | 0
  ACT W: Easy to Wear: 1 | 0 | 0 | 0
  ACT W: Easy to Wear: 2 | 0 | 0 | 1
  ACT W: Easy to Wear: 3 | 5 | 5 | 4
  ACT W: Easy to Wear: 4 | 8 | 9 | 8
  ACT W: Changes the Way I Move: 0 | 0 | 0 | 0
  ACT W: Changes the Way I Move: 1 | 0 | 0 | 0
  ACT W: Changes the Way I Move: 2 | 0 | 0 | 0
  ACT W: Changes the Way I Move: 3 | 4 | 2 | 2
  ACT W: Changes the Way I Move: 4 | 9 | 12 | 11
  ACT W: Changes the Way I Behave: 0 | 0 | 0 | 0
  ACT W: Changes the Way I Behave: 1 | 0 | 1 | 0
  ACT W: Changes the Way I Behave: 2 | 0 | 0 | 0
  ACT W: Changes the Way I Behave: 3 | 5 | 2 | 3
  ACT W: Changes the Way I Behave: 4 | 8 | 11 | 10
  ACT W: Willing to Wear for 4 to 7 Days: 0 | 0 | 0 | 0
  ACT W: Willing to Wear for 4 to 7 Days: 1 | 0 | 0 | 0
  ACT W: Willing to Wear for 4 to 7 Days: 2 | 0 | 0 | 0
  ACT W: Willing to Wear for 4 to 7 Days: 3 | 3 | 5 | 5
  ACT W: Willing to Wear for 4 to 7 Days: 4 | 10 | 9 | 8
  ACT W: Willing to Wear for > 7 Days: 0 | 0 | 0 | 0
  ACT W: Willing to Wear for > 7 Days: 1 | 1 | 0 | 0
  ACT W: Willing to Wear for > 7 Days: 2 | 0 | 0 | 0
  ACT W: Willing to Wear for > 7 Days: 3 | 4 | 5 | 5
  ACT W: Willing to Wear for > 7 Days: 4 | 8 | 9 | 8
  ACT W: If the device could follow my progress during a ttmt, I would wear it: 0 | 0 | 0 | 0
  ACT W: If the device could follow my progress during a ttmt, I would wear it: 1 | 0 | 0 | 0
  ACT W: If the device could follow my progress during a ttmt, I would wear it: 2 | 0 | 0 | 0
  ACT W: If the device could follow my progress during a ttmt, I would wear it: 3 | 4 | 5 | 3
  ACT W: If the device could follow my progress during a ttmt, I would wear it: 4 | 9 | 9 | 10
  ACT W:If device could follow my progress during ttmt, I want my doctor to have access to my results: 0 | 0 | 0 | 0
  ACT W:If device could follow my progress during ttmt, I want my doctor to have access to my results: 1 | 0 | 0 | 0
  ACT W:If device could follow my progress during ttmt, I want my doctor to have access to my results: 2 | 0 | 0 | 0
  ACT W:If device could follow my progress during ttmt, I want my doctor to have access to my results: 3 | 3 | 3 | 4
  ACT W:If device could follow my progress during ttmt, I want my doctor to have access to my results: 4 | 10 | 11 | 9

40. Secondary Outcome: Cohort A: Double Support Duration Measured by ActiGraph and APDM Devices Across Different Floor Surfaces Using Mixed Model Regression Analysis
Description: Double support time referred to the phase during walking when both feet were in contact with the ground. Participants had a single in-lab visit during which they performed gait monitoring procedures. Participants were required to work on tile and carpet at their natural speed while wearing the device under study (ActiGraph) and APDM system. Raw accelerometry data collected by ActiGraph devices was processed by GaitPy to generate gait quality metrics (lumbar position). Gait metrics data was directly extracted from APDM sensors. Analysis was performed using mixed model regression analyses with device, floor type, and their interaction as fixed effects, and participant as random effect.
Time Frame: Up to 20 minutes on Day 1
Population: FAS included all participants who had a signed and dated informed consent document, had assented to the study and were enrolled in the study. The outcome measure was planned to be evaluated only for Cohort A. Mixed model regression analysis did not use age group as a grouping variable and was performed across all participants independent of age groups; hence, combined data is reported for participants aged 3 to 17 years.
Measure: Least Squares Mean (Standard Error); unit: Seconds
Groups:
- Cohort A: Participants Aged 3-17 Years: Participants aged 3 to 17 years wore the ActiGraph CenterPoint Insight Watch on the non-dominant wrist (worn continuously) and lumbar region (worn after waking up in the morning and removed while sleeping at night or nap during daytime) for approximately 15 days (+ 3 days). Participants wore the Ambulatory Parkinson's Disease Monitoring System (APDM) Opal sensors on each wrist, chest, lumbar, and above each shoe, only on Day 1.
Arm/Group | Cohort A: Participants Aged 3-17 Years
Number analyzed (Participants) | 40
Seconds
  ActiGraph: Carpet | 0.28 (0.007)
  APDM: Carpet | 0.20 (0.007)
  ActiGraph: Tile | 0.28 (0.007)
  APDM: Tile | 0.19 (0.007)

41. Secondary Outcome: Cohort A: Single Limb Support Duration Measured by ActiGraph and APDM Devices Across Different Floor Surfaces Using Mixed Model Regression Analysis
Description: Single limb support time referred to the time when only one limb was in contact with the ground. Participants had a single in-lab visit during which they performed gait monitoring procedures. Participants were required to work on tile and carpet at their natural speed while wearing the device under study (ActiGraph) and APDM system. Raw accelerometry data collected by ActiGraph devices was processed by GaitPy to generate gait quality metrics (lumbar position). Gait metrics data was directly extracted from APDM sensors. Analysis was performed using mixed model regression analyses with device, floor type, and their interaction as fixed effects, and participant as random effect.
Time Frame: Up to 20 minutes on Day 1
Population: as for outcome 40
Measure: Least Squares Mean (Standard Error); unit: Seconds
Arm/Group | Cohort A: Participants Aged 3-17 Years
Number analyzed (Participants) | 40
Seconds
  ActiGraph: Carpet | 0.39 (0.006)
  APDM: Carpet | 0.42 (0.006)
  ActiGraph: Tile | 0.38 (0.006)
  APDM: Tile | 0.42 (0.006)

42. Secondary Outcome: Cohort A: Stance Time Measured by ActiGraph and APDM Devices Across Different Floor Surfaces Using Mixed Model Regression Analysis
Description: Stance duration was defined as the duration of time the foot is in contact with the ground in a step during gait. Participants were required to work on tile and carpet at their natural speed while wearing the device under study (ActiGraph) and APDM system. Raw accelerometry data collected by ActiGraph devices was processed by GaitPy to generate gait quality metrics (lumbar position). Gait metrics data was directly extracted from APDM sensors. Analysis was performed using mixed model regression analyses with device, floor type, and their interaction as fixed effects, and participant as random effect.
Time Frame: Up to 20 minutes on Day 1
Population: as for outcome 40
Measure: Least Squares Mean (Standard Error); unit: Seconds
Arm/Group | Cohort A: Participants Aged 3-17 Years
Number analyzed (Participants) | 40
Seconds
  ActiGraph: Carpet | 0.67 (0.012)
  APDM: Carpet | 0.62 (0.012)
  ActiGraph: Tile | 0.66 (0.012)
  APDM: Tile | 0.61 (0.012)

43. Secondary Outcome: Cohort A: Swing Time Measured by ActiGraph and APDM Devices Across Different Floor Surfaces Using Mixed Model Regression Analysis
Description: Swing time was defined as the time during which the foot was not in contact with the ground. Participants were required to work on tile and carpet at their natural speed while wearing the device under study (ActiGraph) and APDM system. Raw accelerometry data collected by ActiGraph devices was processed by GaitPy to generate gait quality metrics (lumbar position). Gait metrics data was directly extracted from APDM sensors. Analysis was performed using mixed model regression analyses with device, floor type, and their interaction as fixed effects, and participant as random effect.
Time Frame: Up to 20 minutes on Day 1
Population: as for outcome 40
Measure: Least Squares Mean (Standard Error); unit: Seconds
Arm/Group | Cohort A: Participants Aged 3-17 Years
Number analyzed (Participants) | 40
Seconds
  ActiGraph: Carpet | 0.39 (0.006)
  APDM: Carpet | 0.42 (0.006)
  ActiGraph: Tile | 0.38 (0.006)
  APDM: Tile | 0.42 (0.006)

44. Secondary Outcome: Cohort A: Stride Length Measured by ActiGraph and APDM Devices Across Different Floor Surfaces Using Mixed Model Regression Analysis
Description: Stride length was defined as the distance covered when two steps were taken, one with each foot. It was measured from the heel of one foot to the heel of same foot when it came into contact with the ground. Participants had a single in-lab visit during which they performed gait monitoring procedures. Participants were required to work on tile and carpet at their natural speed while wearing the device under study (ActiGraph) and APDM system. Raw accelerometry data collected by ActiGraph devices was processed by GaitPy to generate gait quality metrics (lumbar position). Gait metrics data was directly extracted from APDM sensors. Analysis was performed using mixed model regression analyses with device, floor type, and their interaction as fixed effects, and participant as random effect.
Time Frame: Up to 20 minutes on Day 1
Population: as for outcome 40
Measure: Least Squares Mean (Standard Error); unit: Meters
Arm/Group | Cohort A: Participants Aged 3-17 Years
Number analyzed (Participants) | 40
Meters
  ActiGraph: Carpet | 1.00 (0.016)
  APDM: Carpet | 1.01 (0.017)
  ActiGraph: Tile | 1.00 (0.016)
  APDM: Tile | 1.01 (0.016)

45. Secondary Outcome: Cohort A: Step Duration Measured by ActiGraph and APDM Devices Across Different Floor Surfaces Using Mixed Model Regression Analysis
Description: Step duration was the period between the first contact of a foot and the first following contact of the contralateral foot. Participants were required to work on tile and carpet at their natural speed while wearing the device under study (ActiGraph) and APDM system. Raw accelerometry data collected by ActiGraph devices was processed by GaitPy to generate gait quality metrics (lumbar position). Gait metrics data was directly extracted from APDM sensors. Analysis was performed using mixed model regression analyses with device, floor type, and their interaction as fixed effects, and participant as random effect.
Time Frame: Up to 20 minutes on Day 1
Population: as for outcome 40
Measure: Least Squares Mean (Standard Error); unit: Seconds
Arm/Group | Cohort A: Participants Aged 3-17 Years
Number analyzed (Participants) | 40
Seconds
  ActiGraph: Carpet | 0.53 (0.009)
  APDM: Carpet | 0.52 (0.009)
  ActiGraph: Tile | 0.52 (0.009)
  APDM: Tile | 0.51 (0.009)

46. Secondary Outcome: Cohort A: Cadence Measured by ActiGraph and APDM Devices Across Different Floor Surfaces Using Mixed Model Regression Analysis
Description: Cadence referred to the number of steps taken per minute during gait cycle. Participants were required to work on tile and carpet at their natural speed while wearing the device under study (ActiGraph) and APDM system. Raw accelerometry data collected by ActiGraph devices was processed by GaitPy to generate gait quality metrics (lumbar position). Gait metrics data was directly extracted from APDM sensors. Analysis was performed using mixed model regression analyses with device, floor type, and their interaction as fixed effects, and participant as random effect.
Time Frame: Up to 20 minutes on Day 1
Population: as for outcome 40
Measure: Least Squares Mean (Standard Error); unit: Steps per minute
Arm/Group | Cohort A: Participants Aged 3-17 Years
Number analyzed (Participants) | 40
Steps per minute
  ActiGraph: Carpet | 115.08 (2.236)
  APDM: Carpet | 116.79 (2.240)
  ActiGraph: Tile | 117.56 (2.236)
  APDM: Tile | 119.62 (2.236)

47. Secondary Outcome: Cohort A: Gait Speed Measured by ActiGraph and APDM Devices Across Different Floor Surfaces Using Mixed Model Regression Analysis
Description: Gait speed was the time taken to walk a specified distance. Participants were required to work on tile and carpet at their natural speed while wearing the device under study (ActiGraph) and APDM system. Raw accelerometry data collected by ActiGraph devices was processed by GaitPy to generate gait quality metrics (lumbar position). Gait metrics data was directly extracted from APDM sensors. Analysis was performed using mixed model regression analyses with device, floor type, and their interaction as fixed effects, and participant as random effect.
Time Frame: Up to 20 minutes on Day 1
Population: as for outcome 40
Measure: Least Squares Mean (Standard Error); unit: Meters per second
Arm/Group | Cohort A: Participants Aged 3-17 Years
Number analyzed (Participants) | 40
Meters per second
  ActiGraph: Carpet | 0.95 (0.027)
  APDM: Carpet | 0.97 (0.027)
  ActiGraph: Tile | 0.97 (0.027)
  APDM: Tile | 1.00 (0.027)

48. Secondary Outcome: Cohort A: Stride Duration Measured by ActiGraph and APDM Devices Across Different Floor Surfaces Using Mixed Model Regression Analysis
Description: Stride duration refers to the duration between successive heel contacts of the same foot. Participants were required to work on tile and carpet at their natural speed while wearing the device under study (ActiGraph) and APDM system. Raw accelerometry data collected by ActiGraph devices was processed by GaitPy to generate gait quality metrics (lumbar position). Gait metrics data was directly extracted from APDM sensors. Analysis was performed using mixed model regression analyses with device, floor type, and their interaction as fixed effects, and participant as random effect.
Time Frame: Up to 20 minutes on Day 1
Population: as for outcome 40
Measure: Least Squares Mean (Standard Error); unit: Seconds
Arm/Group | Cohort A: Participants Aged 3-17 Years
Number analyzed (Participants) | 40
Seconds
  ActiGraph: Carpet | 1.05 (0.018)
  APDM: Carpet | 1.04 (0.018)
  ActiGraph: Tile | 1.04 (0.018)
  APDM: Tile | 1.02 (0.018)

49. Secondary Outcome: Cohort B: Number of Hours Per Day Wearing the Panoramic Bracelet Devices at Home
Time Frame: From Day 1 up to Day 7
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: Hours per day
Arm/Group | Cohort B: Participants Aged 3-5 Years | Cohort B: Participants Aged 6-11 Years | Cohort B: Participants Aged 12-17 Years
Number analyzed (Participants) | 13 | 17 | 17
Hours per day | 22.65 (1.051) | 22.80 (1.317) | 22.60 (1.590)

50. Secondary Outcome: Cohort B: Double Support Duration Measured by APDM, GAITRite Walkway and Panoramic Bracelet Devices for Walk at Natural, Slow and Fast Speed Tasks
Description: Double support time referred to the phase during walking when both feet were in contact with the ground. Participants had to walk on GAITRite walkway (20 feet*3) wearing Panoramic bracelet device and APDM devices at participant's natural speed and at varied speeds. Natural speed was participant's self-chosen pace for 3 rounds. Varied speeds included participant's self-chosen slow pace ("Walk slow") and fast pace ("Walk fast") for 3 rounds. Raw accelerometry data collected by devices were processed by manufacturer's algorithm for APDM and SKDH gait algorithm for Panoramic bracelet device to generate gait metrics.
Time Frame: Up to 20 minutes on Day 1
Population: FAS included all participants who had a signed and dated informed consent document, had assented to the study and were enrolled in the study. Here, 'Number Analyzed' signifies number of participants evaluable for the specified rows. The outcome measure was planned to be evaluated only for Cohort B.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Cohort B: Participants Aged 3-5 Years | Cohort B: Participants Aged 6-11 Years | Cohort B: Participants Aged 12-17 Years
Number analyzed (Participants) | 13 | 17 | 17
Seconds
  Panoramic Bracelet: Natural Speed | 0.29 (0.063) | 0.32 (0.031) | 0.34 (0.035)
  GAITRite: Natural Speed | 0.20 (0.038) | 0.25 (0.041) | 0.31 (0.032)
  APDM: Natural Speed: number analyzed (Participants) | 11 | 17 | 17
  APDM: Natural Speed | 0.16 (0.031) | 0.17 (0.039) | 0.19 (0.041)
  Panoramic Bracelet: Fast Speed: number analyzed (Participants) | 12 | 17 | 17
  Panoramic Bracelet: Fast Speed | 0.24 (0.056) | 0.26 (0.047) | 0.30 (0.030)
  GAITRite: Fast Speed: number analyzed (Participants) | 12 | 17 | 17
  GAITRite: Fast Speed | 0.15 (0.040) | 0.18 (0.041) | 0.24 (0.030)
  APDM: Fast Speed: number analyzed (Participants) | 5 | 14 | 16
  APDM: Fast Speed | 0.13 (0.032) | 0.12 (0.027) | 0.15 (0.031)
  Panoramic Bracelet: Slow Speed: number analyzed (Participants) | 12 | 17 | 17
  Panoramic Bracelet: Slow Speed | 0.42 (0.166) | 0.50 (0.183) | 0.51 (0.121)
  GAITRite: Slow Speed: number analyzed (Participants) | 12 | 17 | 17
  GAITRite: Slow Speed | 0.37 (0.181) | 0.47 (0.243) | 0.52 (0.148)
  APDM: Slow Speed: number analyzed (Participants) | 11 | 17 | 17
  APDM: Slow Speed | 0.34 (0.179) | 0.37 (0.199) | 0.37 (0.122)

51. Secondary Outcome: Cohort B: Single Limb Support Duration Measured by APDM, GAITRite Walkway and Panoramic Bracelet Devices for Walk at Natural, Slow and Fast Speed Tasks
Description: Single support time referred to the time when only one limb was in contact with the ground. Participants had to walk on GAITRite walkway (20 feet*3) wearing Panoramic bracelet device and APDM devices at participant's natural speed and at varied speeds. Natural speed was participant's self-chosen pace for 3 rounds. Varied speeds included participant's self-chosen slow pace ("Walk slow") and fast pace ("Walk fast") for 3 rounds. Raw accelerometry data collected by devices were processed by manufacturer's algorithm for APDM and SKDH gait algorithm for Panoramic bracelet device to generate gait metrics.
Time Frame: Up to 20 minutes on Day 1
Population: as for outcome 50
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Cohort B: Participants Aged 3-5 Years | Cohort B: Participants Aged 6-11 Years | Cohort B: Participants Aged 12-17 Years
Number analyzed (Participants) | 13 | 17 | 17
Seconds
  Panoramic Bracelet: Natural Speed | 0.31 (0.111) | 0.34 (0.036) | 0.39 (0.026)
  GAITRite: Natural Speed | 0.31 (0.016) | 0.37 (0.031) | 0.39 (0.027)
  APDM: Natural Speed: number analyzed (Participants) | 11 | 17 | 17
  APDM: Natural Speed | 0.36 (0.021) | 0.41 (0.034) | 0.45 (0.027)
  Panoramic Bracelet: Fast Speed: number analyzed (Participants) | 12 | 17 | 17
  Panoramic Bracelet: Fast Speed | 0.26 (0.052) | 0.29 (0.029) | 0.35 (0.029)
  GAITRite: Fast Speed: number analyzed (Participants) | 12 | 17 | 17
  GAITRite: Fast Speed | 0.30 (0.027) | 0.32 (0.030) | 0.37 (0.025)
  APDM: Fast Speed: number analyzed (Participants) | 5 | 15 | 16
  APDM: Fast Speed | 0.34 (0.018) | 0.37 (0.031) | 0.42 (0.028)
  Panoramic Bracelet: Slow Speed: number analyzed (Participants) | 12 | 17 | 17
  Panoramic Bracelet: Slow Speed | 0.50 (0.356) | 0.48 (0.140) | 0.51 (0.102)
  GAITRite: Slow Speed: number analyzed (Participants) | 12 | 17 | 17
  GAITRite: Slow Speed | 0.36 (0.079) | 0.46 (0.141) | 0.50 (0.095)
  APDM: Slow Speed: number analyzed (Participants) | 11 | 17 | 17
  APDM: Slow Speed | 0.43 (0.088) | 0.52 (0.151) | 0.58 (0.112)

52. Secondary Outcome: Cohort B: Stance Duration Measured by APDM, GAITRite Walkway and Panoramic Bracelet Devices for Walk at Natural, Slow and Fast Speed Tasks
Description: Stance duration was defined as the duration of time the foot is in contact with the ground in a step during gait. Participants had to walk on GAITRite walkway (20 feet*3) wearing Panoramic bracelet device and APDM devices at participant's natural speed and at varied speeds. Natural speed was participant's self-chosen pace for 3 rounds. Varied speeds included participant's self-chosen slow pace ("Walk slow") and fast pace ("Walk fast") for 3 rounds. Raw accelerometry data collected by devices were processed by manufacturer's algorithm for APDM and SKDH gait algorithm for Panoramic bracelet device to generate gait metrics.
Time Frame: Up to 20 minutes on Day 1
Population: as for outcome 50
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Cohort B: Participants Aged 3-5 Years | Cohort B: Participants Aged 6-11 Years | Cohort B: Participants Aged 12-17 Years
Number analyzed (Participants) | 13 | 17 | 17
Seconds
  Panoramic Bracelet: Natural Speed | 0.61 (0.186) | 0.66 (0.062) | 0.73 (0.055)
  GAITRite: Natural Speed | 0.52 (0.048) | 0.63 (0.064) | 0.71 (0.051)
  APDM: Natural Speed: number analyzed (Participants) | 11 | 17 | 17
  APDM: Natural Speed | 0.52 (0.044) | 0.58 (0.061) | 0.64 (0.054)
  Panoramic Bracelet: Fast Speed: number analyzed (Participants) | 12 | 17 | 17
  Panoramic Bracelet: Fast Speed | 0.52 (0.100) | 0.55 (0.069) | 0.64 (0.048)
  GAITRite: Fast Speed: number analyzed (Participants) | 12 | 17 | 17
  GAITRite: Fast Speed | 0.44 (0.063) | 0.51 (0.064) | 0.62 (0.050)
  APDM: Fast Speed: number analyzed (Participants) | 5 | 15 | 16
  APDM: Fast Speed | 0.47 (0.037) | 0.48 (0.050) | 0.56 (0.044)
  Panoramic Bracelet: Slow Speed: number analyzed (Participants) | 12 | 17 | 17
  Panoramic Bracelet: Slow Speed | 0.91 (0.452) | 0.99 (0.340) | 1.03 (0.230)
  GAITRite: Slow Speed: number analyzed (Participants) | 12 | 17 | 17
  GAITRite: Slow Speed | 0.74 (0.245) | 0.93 (0.342) | 1.03 (0.232)
  APDM: Slow Speed: number analyzed (Participants) | 11 | 17 | 17
  APDM: Slow Speed | 0.78 (0.256) | 0.89 (0.352) | 0.95 (0.228)

53. Secondary Outcome: Cohort B: Swing Duration Measured by APDM, GAITRite Walkway and Panoramic Bracelet Devices for Walk at Natural, Slow and Fast Speed Tasks
Description: Swing time was defined as the time during which the foot was not in contact with the ground. Participants had to walk on GAITRite walkway (20 feet*3) wearing Panoramic bracelet device and APDM devices at participant's natural speed and at varied speeds. Natural speed was participant's self-chosen pace for 3 rounds. Varied speeds included participant's self-chosen slow pace ("Walk slow") and fast pace ("Walk fast") for 3 rounds. Raw accelerometry data collected by devices were processed by manufacturer's algorithm for APDM and SKDH gait algorithm for Panoramic bracelet device to generate gait metrics.
Time Frame: Up to 20 minutes on Day 1
Population: as for outcome 50
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Cohort B: Participants Aged 3-5 Years | Cohort B: Participants Aged 6-11 Years | Cohort B: Participants Aged 12-17 Years
Number analyzed (Participants) | 13 | 17 | 17
Seconds
  Panoramic Bracelet: Natural Speed | 0.30 (0.085) | 0.34 (0.036) | 0.38 (0.026)
  GAITRite: Natural Speed | 0.32 (0.016) | 0.37 (0.032) | 0.39 (0.026)
  APDM: Natural Speed: number analyzed (Participants) | 11 | 17 | 17
  APDM: Natural Speed | 0.36 (0.015) | 0.41 (0.034) | 0.45 (0.027)
  Panoramic Bracelet: Fast Speed: number analyzed (Participants) | 12 | 17 | 17
  Panoramic Bracelet: Fast Speed | 0.26 (0.051) | 0.29 (0.029) | 0.34 (0.029)
  GAITRite: Fast Speed: number analyzed (Participants) | 12 | 17 | 17
  GAITRite: Fast Speed | 0.30 (0.026) | 0.33 (0.029) | 0.37 (0.026)
  APDM: Fast Speed: number analyzed (Participants) | 5 | 15 | 16
  APDM: Fast Speed | 0.34 (0.017) | 0.37 (0.031) | 0.42 (0.026)
  Panoramic Bracelet: Slow Speed: number analyzed (Participants) | 11 | 17 | 17
  Panoramic Bracelet: Slow Speed | 0.39 (0.182) | 0.48 (0.137) | 0.51 (0.102)
  GAITRite: Slow Speed: number analyzed (Participants) | 11 | 17 | 17
  GAITRite: Slow Speed | 0.36 (0.081) | 0.46 (0.139) | 0.50 (0.095)
  APDM: Slow Speed: number analyzed (Participants) | 12 | 17 | 17
  APDM: Slow Speed | 0.43 (0.087) | 0.52 (0.140) | 0.57 (0.109)

54. Secondary Outcome: Cohort B: Stride Length Measured by APDM, GAITRite Walkway and Panoramic Bracelet Devices for Walk at Natural, Slow and Fast Speed Tasks
Description: Stride length was defined as the distance covered when two steps were taken, one with each foot. It was measured from the heel of one foot to the heel of same foot when it came into contact with the ground. Participants had to walk on GAITRite walkway (20 feet*3) wearing Panoramic bracelet device and APDM devices at participant's natural speed and at varied speeds. Natural speed was participant's self-chosen pace for 3 rounds. Varied speeds included participant's self-chosen slow pace ("Walk slow") and fast pace ("Walk fast") for 3 rounds. Raw accelerometry data collected by devices were processed by manufacturer's algorithm for APDM and SKDH gait algorithm for Panoramic bracelet device to generate gait metrics.
Time Frame: Up to 20 minutes on Day 1
Population: as for outcome 50
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Cohort B: Participants Aged 3-5 Years | Cohort B: Participants Aged 6-11 Years | Cohort B: Participants Aged 12-17 Years
Number analyzed (Participants) | 13 | 17 | 17
Meters
  Panoramic Bracelet: Natural Speed | 1.01 (0.182) | 1.24 (0.166) | 1.29 (0.149)
  GAITRite: Natural Speed | 0.88 (0.122) | 1.20 (0.093) | 1.37 (0.094)
  APDM: Natural Speed: number analyzed (Participants) | 11 | 17 | 17
  APDM: Natural Speed | 0.78 (0.104) | 1.09 (0.091) | 1.23 (0.093)
  Panoramic Bracelet: Fast Speed: number analyzed (Participants) | 12 | 17 | 17
  Panoramic Bracelet: Fast Speed | 1.17 (0.320) | 1.33 (0.163) | 1.48 (0.197)
  GAITRite: Fast Speed: number analyzed (Participants) | 12 | 17 | 17
  GAITRite: Fast Speed | 1.02 (0.101) | 1.34 (0.106) | 1.56 (0.159)
  APDM: Fast Speed: number analyzed (Participants) | 5 | 15 | 16
  APDM: Fast Speed | 0.88 (0.073) | 1.23 (0.109) | 1.39 (0.120)
  Panoramic Bracelet: Slow Speed: number analyzed (Participants) | 11 | 17 | 17
  Panoramic Bracelet: Slow Speed | 0.85 (0.211) | 0.99 (0.244) | 1.06 (0.127)
  GAITRite: Slow Speed: number analyzed (Participants) | 11 | 17 | 17
  GAITRite: Slow Speed | 0.61 (0.174) | 0.90 (0.217) | 1.11 (0.122)
  APDM: Slow Speed: number analyzed (Participants) | 12 | 17 | 17
  APDM: Slow Speed | 0.51 (0.157) | 0.78 (0.194) | 0.94 (0.112)

55. Secondary Outcome: Cohort B: Step Duration Measured by APDM, GAITRite Walkway and Panoramic Bracelet Devices for Walk at Natural, Slow and Fast Speed Tasks
Description: Step duration was the period between the first contact of a foot and the first following contact of the contralateral foot. Participants had to walk on GAITRite walkway (20 feet*3) wearing Panoramic bracelet device and APDM devices at participant's natural speed and at varied speeds. Natural speed was participant's self-chosen pace for 3 rounds. Varied speeds included participant's self-chosen slow pace ("Walk slow") and fast pace ("Walk fast") for 3 rounds. Raw accelerometry data collected by devices were processed by manufacturer's algorithm for APDM and SKDH gait algorithm for Panoramic bracelet device to generate gait metrics.
Time Frame: Up to 20 minutes on Day 1
Population: as for outcome 50
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Cohort B: Participants Aged 3-5 Years | Cohort B: Participants Aged 6-11 Years | Cohort B: Participants Aged 12-17 Years
Number analyzed (Participants) | 13 | 17 | 17
Seconds
  Panoramic Bracelet: Natural Speed | 0.46 (0.152) | 0.50 (0.046) | 0.55 (0.037)
  GAITRite: Natural Speed | 0.42 (0.030) | 0.49 (0.044) | 0.55 (0.037)
  APDM: Natural Speed: number analyzed (Participants) | 11 | 17 | 17
  APDM: Natural Speed | 0.44 (0.024) | 0.50 (0.046) | 0.55 (0.037)
  Panoramic Bracelet: Fast Speed: number analyzed (Participants) | 12 | 17 | 17
  Panoramic Bracelet: Fast Speed | 0.39 (0.074) | 0.42 (0.042) | 0.50 (0.038)
  GAITRite: Fast Speed: number analyzed (Participants) | 12 | 17 | 17
  GAITRite: Fast Speed | 0.37 (0.044) | 0.42 (0.047) | 0.49 (0.036)
  APDM: Fast Speed: number analyzed (Participants) | 5 | 15 | 16
  APDM: Fast Speed | 0.40 (0.026) | 0.43 (0.042) | 0.49 (0.033)
  Panoramic Bracelet: Slow Speed: number analyzed (Participants) | 12 | 17 | 17
  Panoramic Bracelet: Slow Speed | 0.70 (0.418) | 0.74 (0.241) | 0.77 (0.164)
  GAITRite: Slow Speed: number analyzed (Participants) | 12 | 17 | 17
  GAITRite: Slow Speed | 0.54 (0.157) | 0.70 (0.229) | 0.76 (0.165)
  APDM: Slow Speed: number analyzed (Participants) | 11 | 17 | 17
  APDM: Slow Speed | 0.60 (0.171) | 0.71 (0.247) | 0.76 (0.162)

56. Secondary Outcome: Cohort B: Cadence Measured by APDM, GAITRite Walkway and Panoramic Bracelet Devices for Walk at Natural, Slow and Fast Speed Tasks
Description: Cadence referred to the number of steps taken per minute during gait cycle. Participants had to walk on GAITRite walkway (20 feet*3) wearing Panoramic bracelet device and APDM devices at participant's natural speed and at varied speeds. Natural speed was participant's self-chosen pace for 3 rounds. Varied speeds included participant's self-chosen slow pace ("Walk slow") and fast pace ("Walk fast") for 3 rounds. Raw accelerometry data collected by devices were processed by manufacturer's algorithm for APDM and SKDH gait algorithm for Panoramic bracelet device to generate gait metrics.
Time Frame: Up to 20 minutes on Day 1
Population: as for outcome 50
Measure: Mean (Standard Deviation); unit: Steps per minute
Arm/Group | Cohort B: Participants Aged 3-5 Years | Cohort B: Participants Aged 6-11 Years | Cohort B: Participants Aged 12-17 Years
Number analyzed (Participants) | 13 | 17 | 17
Steps per minute
  Panoramic Bracelet: Natural Speed | 138.45 (26.272) | 119.94 (10.909) | 108.89 (7.163)
  GAITRite: Natural Speed | 144.80 (11.373) | 122.16 (10.433) | 109.98 (7.504)
  APDM: Natural Speed: number analyzed (Participants) | 11 | 17 | 17
  APDM: Natural Speed | 136.44 (7.962) | 122.15 (10.904) | 110.45 (7.473)
  Panoramic Bracelet: Fast Speed: number analyzed (Participants) | 12 | 17 | 17
  Panoramic Bracelet: Fast Speed | 158.13 (28.017) | 144.41 (14.793) | 121.24 (9.227)
  GAITRite: Fast Speed: number analyzed (Participants) | 12 | 17 | 17
  GAITRite: Fast Speed | 166.43 (20.297) | 145.96 (16.900) | 122.86 (9.042)
  APDM: Fast Speed: number analyzed (Participants) | 5 | 15 | 16
  APDM: Fast Speed | 147.01 (11.303) | 141.76 (13.502) | 122.66 (8.589)
  Panoramic Bracelet: Slow Speed: number analyzed (Participants) | 12 | 17 | 17
  Panoramic Bracelet: Slow Speed | 106.99 (45.694) | 88.81 (24.208) | 81.21 (16.065)
  GAITRite: Slow Speed: number analyzed (Participants) | 12 | 17 | 17
  GAITRite: Slow Speed | 119.25 (36.642) | 93.91 (25.728) | 82.24 (16.459)
  APDM: Slow Speed: number analyzed (Participants) | 11 | 17 | 17
  APDM: Slow Speed | 106.81 (28.903) | 92.80 (25.727) | 82.07 (16.271)

57. Secondary Outcome: Cohort B: Gait Speed Measured by APDM, GAITRite Walkway and Panoramic Bracelet Devices for Walk at Natural, Slow and Fast Speed Task
Description: Gait speed was the time taken to walk a specified distance. Participants had to walk on GAITRite walkway (20 feet*3) wearing Panoramic bracelet device and APDM devices at participant's natural speed and at varied speeds. Natural speed was participant's self-chosen pace for 3 rounds. Varied speeds included participant's self-chosen slow pace ("Walk slow") and fast pace ("Walk fast") for 3 rounds. Raw accelerometry data collected by devices were processed by manufacturer's algorithm for APDM and SKDH gait algorithm for Panoramic bracelet device to generate gait metrics.
Time Frame: Up to 20 minutes on Day 1
Population: as for outcome 50
Measure: Mean (Standard Deviation); unit: Meters per second
Arm/Group | Cohort B: Participants Aged 3-5 Years | Cohort B: Participants Aged 6-11 Years | Cohort B: Participants Aged 12-17 Years
Number analyzed (Participants) | 13 | 17 | 17
Meters per second
  Panoramic Bracelet: Natural Speed | 1.15 (0.209) | 1.24 (0.228) | 1.17 (0.176)
  GAITRite: Natural Speed | 1.07 (0.211) | 1.21 (0.144) | 1.25 (0.124)
  APDM: Natural Speed: number analyzed (Participants) | 11 | 17 | 17
  APDM: Natural Speed | 0.89 (0.147) | 1.11 (0.144) | 1.13 (0.120)
  Panoramic Bracelet: Fast Speed: number analyzed (Participants) | 12 | 17 | 17
  Panoramic Bracelet: Fast Speed | 1.50 (0.345) | 1.57 (0.191) | 1.50 (0.262)
  GAITRite: Fast Speed: number analyzed (Participants) | 12 | 17 | 17
  GAITRite: Fast Speed | 1.41 (0.234) | 1.63 (0.205) | 1.59 (0.225)
  APDM: Fast Speed: number analyzed (Participants) | 5 | 15 | 16
  APDM: Fast Speed | 1.07 (0.105) | 1.45 (0.130) | 1.43 (0.162)
  Panoramic Bracelet: Slow Speed: number analyzed (Participants) | 11 | 17 | 17
  Panoramic Bracelet: Slow Speed | 0.77 (0.298) | 0.72 (0.223) | 0.73 (0.171)
  GAITRite: Slow Speed: number analyzed (Participants) | 12 | 17 | 17
  GAITRite: Slow Speed | 0.59 (0.256) | 0.70 (0.280) | 0.76 (0.174)
  APDM: Slow Speed: number analyzed (Participants) | 11 | 17 | 17
  APDM: Slow Speed | 0.47 (0.224) | 0.61 (0.273) | 0.65 (0.168)

58. Secondary Outcome: Cohort B: Stride Duration Measured by APDM, GAITRite Walkway and Panoramic Bracelet Devices for Walk at Natural, Slow and Fast Speed Tasks
Description: Stride duration refers to the duration between successive heel contacts of the same foot. Participants had to walk on GAITRite walkway (20 feet*3) wearing Panoramic bracelet device and APDM devices at participant's natural speed and at varied speeds. Natural speed was participant's self-chosen pace for 3 rounds. Varied speeds included participant's self-chosen slow pace ("Walk slow") and fast pace ("Walk fast") for 3 rounds. Raw accelerometry data collected by devices were processed by manufacturer's algorithm for APDM and SKDH gait algorithm for Panoramic bracelet device to generate gait metrics.
Time Frame: Up to 20 minutes on Day 1
Population: as for outcome 50
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Cohort B: Participants Aged 3-5 Years | Cohort B: Participants Aged 6-11 Years | Cohort B: Participants Aged 12-17 Years
Number analyzed (Participants) | 13 | 17 | 17
Seconds
  Panoramic Bracelet: Natural Speed | 0.90 (0.257) | 1.00 (0.093) | 1.11 (0.078)
  GAITRite: Natural Speed | 0.84 (0.070) | 0.99 (0.091) | 1.10 (0.073)
  APDM: Natural Speed: number analyzed (Participants) | 11 | 17 | 17
  APDM: Natural Speed | 0.88 (0.055) | 0.99 (0.093) | 1.09 (0.074)
  Panoramic Bracelet: Fast Speed: number analyzed (Participants) | 12 | 17 | 17
  Panoramic Bracelet: Fast Speed | 0.78 (0.140) | 0.84 (0.093) | 0.99 (0.075)
  GAITRite: Fast Speed: number analyzed (Participants) | 12 | 17 | 17
  GAITRite: Fast Speed | 0.73 (0.085) | 0.83 (0.094) | 0.98 (0.071)
  APDM: Fast Speed: number analyzed (Participants) | 5 | 15 | 16
  APDM: Fast Speed | 0.82 (0.063) | 0.85 (0.079) | 0.98 (0.069)
  Panoramic Bracelet: Slow Speed: number analyzed (Participants) | 11 | 17 | 17
  Panoramic Bracelet: Slow Speed | 1.24 (0.552) | 1.46 (0.477) | 1.53 (0.326)
  GAITRite: Slow Speed: number analyzed (Participants) | 12 | 17 | 17
  GAITRite: Slow Speed | 1.12 (0.352) | 1.40 (0.473) | 1.52 (0.330)
  APDM: Slow Speed: number analyzed (Participants) | 11 | 17 | 17
  APDM: Slow Speed | 1.20 (0.336) | 1.42 (0.489) | 1.52 (0.330)

ADVERSE EVENTS:
Time Frame: From Day 1 to Day 15 (+3 days)
Description: FAS included all participants who had a signed and dated informed consent document, had assented to the study and were enrolled in the study.
Arm/Group | Cohort A: Participants Aged 3-5 Years | Cohort A: Participants Aged 6-11 Years | Cohort A: Participants Aged 12-17 Years | Cohort B: Participants Aged 3-5 Years | Cohort B: Participants Aged 6-11 Years | Cohort B: Participants Aged 12-17 Years
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/14 | 0/13 | 0/13 | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/14 | 0/13 | 0/13 | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 4/13 | 3/14 | 3/13 | 2/13 | 4/17 | 3/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: Participants Aged 3-5 Years (N=13) | Cohort A: Participants Aged 6-11 Years (N=14) | Cohort A: Participants Aged 12-17 Years (N=13) | Cohort B: Participants Aged 3-5 Years (N=13) | Cohort B: Participants Aged 6-11 Years (N=17) | Cohort B: Participants Aged 12-17 Years (N=17)
Medical device site bruise (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 — MedDRA 25.1 for Cohort A and MedDRA 27.1 for Cohort B
Pyrexia (General disorders) | 0 | 1 | 1 | 0 | 1 | 0 — MedDRA 25.1 for Cohort A and MedDRA 27.1 for Cohort B
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 — MedDRA 25.1 for Cohort A and MedDRA 27.1 for Cohort B
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 — MedDRA 25.1 for Cohort A and MedDRA 27.1 for Cohort B
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA 25.1 for Cohort A and MedDRA 27.1 for Cohort B
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA 25.1 for Cohort A and MedDRA 27.1 for Cohort B
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 — MedDRA 25.1 for Cohort A and MedDRA 27.1 for Cohort B
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA 25.1 for Cohort A and MedDRA 27.1 for Cohort B
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 2 | 1 — MedDRA 25.1 for Cohort A and MedDRA 27.1 for Cohort B
Skin indentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 — MedDRA 25.1 for Cohort A and MedDRA 27.1 for Cohort B
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 — MedDRA 25.1 for Cohort A and MedDRA 27.1 for Cohort B
Medical device site irritation (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA 25.1 for Cohort A and MedDRA 27.1 for Cohort B
Medical device site rash (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA 25.1 for Cohort A and MedDRA 27.1 for Cohort B
Upper respiratory tract infection (Infections and infestations) | 3 | 0 | 0 | 0 | 0 | 0 — MedDRA 25.1 for Cohort A and MedDRA 27.1 for Cohort B
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA 25.1 for Cohort A and MedDRA 27.1 for Cohort B
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 — MedDRA 25.1 for Cohort A and MedDRA 27.1 for Cohort B

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2023-04-12): https://cdn.clinicaltrials.gov/large-docs/50/NCT04823650/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-06): https://cdn.clinicaltrials.gov/large-docs/50/NCT04823650/SAP_001.pdf